CLINICAL TRIAL: NCT03633227
Title: A Phase 4, Double-Blind, Randomized, Placebo-Controlled Study Evaluating the Pharmacokinetics and Safety of Obeticholic Acid in Patients With Primary Biliary Cholangitis and Moderate to Severe Hepatic Impairment
Brief Title: Study of Obeticholic Acid (OCA) Evaluating Pharmacokinetics and Safety in Participants With Primary Biliary Cholangitis (PBC) and Hepatic Impairment
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to Ocaliva (obeticholic acid) US labeling update, the sponsor decided to terminate the study.
Sponsor: Intercept Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 747-401
Record Dates: First submitted 2018-04-08; First posted 2018-08-16 (Actual); Results first posted 2022-09-06 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-08

CONDITIONS: Liver Cirrhosis, Biliary
Keywords: Primary Biliary Cholangitis; Primary Biliary Cirrhosis; PBC; Hepatic Impairment; Cirrhosis; Liver
MeSH Terms: conditions — Liver Cirrhosis, Biliary; Fibrosis | interventions — obeticholic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Obeticholic Acid (OCA) (Experimental): Participants will initiate treatment with OCA 5 milligrams (mg) tablets orally once weekly. At Week 12, if there are no safety concerns, the dose will be up-titrated to OCA 5 mg twice weekly. Every 6 weeks thereafter, based on tolerability assessments, further up-titration of dose will be considered. At each titration visit, the participants will start the higher dose regimen no earlier than 2 days after the prior dose. The maximum dose titration will be OCA 10 mg twice weekly at least 3 days apart. The minimum treatment duration will be 48-weeks. Participants, who complete their 48-week treatment, can continue the treatment until all randomized participants complete their 48-week treatment period and the database for that period is locked (total duration: approximately up to 3 years).
  Interventions: Drug: Obeticholic Acid (OCA)
- Placebo (Placebo Comparator): Participants will receive OCA matching placebo orally once weekly or twice weekly for the duration of at least 48-weeks. Participants, who complete their 48-week treatment, can continue the treatment until all randomized participants complete their 48-week treatment period and the database for that period is locked (total duration: approximately up to 3 years).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Obeticholic Acid (OCA) — OCA will be administered per dose and schedule specified in the arm description.
  Other Names: 6alpha-ethylchenodeoxycholic acid (6-ECDCA); INT-747
  Arms: Obeticholic Acid (OCA)
Drug: Placebo — OCA matching placebo will be administered per the schedule specified in the arm description.
  Arms: Placebo

SUMMARY:
This Phase 4, randomized, double-blind, placebo-controlled study will evaluate the pharmacokinetics (PK) and safety of OCA treatment in participants with PBC and moderate to severe hepatic impairment over a 48-week treatment period. Participants who have completed their 48-week double blind treatment period will continue double-blind treatment until all randomized participants have completed their 48-week treatment period and the database for that period is locked. An open-label extension study in which all participants receive OCA will be considered following review of blinded safety and PK data.

ELIGIBILITY:
Inclusion Criteria:

1. A definite or probable diagnosis of PBC (consistent with American Association for the Study of Liver Diseases [AASLD] and European Association for the Study of the Liver [EASL] Practice Guidelines, defined as having ≥2 of the following 3 diagnostic factors:

   * History of elevated alkaline phosphatase (ALP) levels for at least 6 months
   * Positive antimitochondrial antibody (AMA) titer or if AMA negative or low titer (≤1:80), PBC specific antibodies (anti-glycoprotein 210 [GP210] and/or anti-SP100) and/or antibodies against the major M2 components (E2 component of mitochondrial pyruvate dehydrogenase complex [PDC-E2], 2-oxo-glutaric acid dehydrogenase complex)
   * Liver biopsy consistent with PBC (collected at any time prior to Screening)
2. Evidence of cirrhosis including at least one of the following:

   * Biopsy results consistent with PBC Stage 4
   * Liver stiffness as assessed by Transient Elastography (TE) Median Value ≥16.9 kilopascals (kPa)
   * Clinical evidence in the absence of acute liver failure consistent with cirrhosis including: gastroesophageal varices, ascites, radiological evidence of cirrhosis (nodular liver or enlargement of portal vein and splenomegaly)
   * Combined low platelet count (<140,000/cubic millimeter [mm^3]) with

     * persistent decrease in serum albumin, or
     * elevation in prothrombin time/international normalized ratio (INR) (not due to antithrombotic agent use), or
     * elevated bilirubin (2*upper limit of normal [ULN])
3. Satisfy the criteria of the modified Child-Pugh (CP) classification for hepatic impairment during Screening:

   * Moderate: CP-B (Scores 7 to 9) or
   * Severe: CP-C (Scores 10 to 12)
4. Model of end-stage liver disease (MELD) score of 6 to 24 at Screening
5. Taking ursodeoxycholic acid (UDCA) for at least 12 months (stable dose for ≥3 months) prior to Day 1, or unable to tolerate or unresponsive to UDCA (no UDCA for ≥3 months)

Exclusion Criteria:

1. Non-cirrhotic or cirrhotic CP-A (Mild; Score 5 to 6)
2. History of liver transplant or organ transplant
3. History of alcohol or drug abuse within 12 months prior to Screening
4. Hepatic encephalopathy (as defined by a West Haven score of ≥2
5. History or presence of other concomitant liver diseases including:

   * Hepatitis C virus infection and ribonucleic acid (RNA) positive
   * Active hepatitis B infection; however, participants who have seroconverted (hepatitis B surface antigen and hepatitis B e antigen negative) may be included in this study after consultation with the medical monitor
   * Primary sclerosing cholangitis
   * Alcoholic liver disease
   * Definite autoimmune liver disease or overlap hepatitis
   * Gilbert's Syndrome
6. In the opinion of the Investigator, fluctuating or rapidly deteriorating hepatic function prior to randomization

Other inclusion/exclusion criteria may apply.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-06-22 (Actual); Primary Completion 2021-07-09 (Actual); Study Completion 2021-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Shiff, M.D., Study Director — Intercept Pharmaceuticals
Locations (40):
- United States (11):
  - Inland Empire Liver Foundation, Rialto, California
  - University of California, Ddavis Medical Center, Sacramento, California
  - Schiff Center for Liver Diseases/ University of Miami, Miami, Florida
  - Mercy Medical Center, Baltimore, Maryland
  - University Of Michigan, Ann Arbor, Michigan
  - Kansas City Research Institute, Kansas City, Missouri
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - UPMC Center for Liver Diseases, Pittsburgh, Pennsylvania
  - The Liver Institute at Methodist Dallas Medical Center, Dallas, Texas
  - Baylor College of Medicine- Advanced Liver Therapies, Houston, Texas
  - American Research Corporation at theTexas Liver Institute, San Antonio, Texas
- Argentina (8):
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Hospital Universitario Austral, Buenos Aires
  - Hospital Aleman, Caba
  - Hospital Britanico de Buenos Aires, Caba
  - Hospital de Gastroenterologia "Dr Carlos Bonorino Udaondo", Ciudad Autonoma de Buenos Aire
  - Higea S.A., Mendoza
  - Hospital Universitario Austral, Pilar
  - Hospital Provincial del Centenario, Rosario
- Australia (2):
  - Royal Prince Alfred Hospital, Camperdown
  - Nepean Hospital, Kingswood
- Belgium (3):
  - CUB Hospital Erasme, Brussels
  - Universitair Ziekenhuis Antwerpen UZA, Edegem
  - University Hospital Leuven, Leuven
- Brazil (3):
  - Hospital das Clínicas da Universidade Federal de Minas Gerais - UFMG, Belo Horizonte
  - Hospital de Clinicas de Porto Alegre, Rio Grande
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo
- Toronto General Hospital, Toronto, Canada
- Estonia (2):
  - West Tallinn Central Hospital, Tallinn
  - Tartu University Hospital, Tartu
- Universitatsklinikum Leipzig AoR, Leipzig, Germany
- Bekes Megyei Kozponti Korhaz Dr. Rethy Pal Tagkorhaz, 4. Belgyogyaszat-Gasztroenterologia-Hepatologia, Békéscsaba, Hungary
- Italy (2):
  - Azienda Socio Sanitaria Territoriale (ASST) di Monza, Monza, MB
  - AOU Ospedale Civile S. Agostino Estense - UO Medicina Metabolica, Modena
- Lithuania (3):
  - Hospital of Lithuanian University of Health Sciences Kauno Klinikos, Kaunas
  - Klaipeda Seamen's Hospital, Klaipėda
  - Vilnius University Hospital Santaros Klinikos, Vilnius
- Spain (3):
  - Paseo Vall d'Hebron, Barcelona
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitari I Politecnic La Fe de Valencia, Valencia

REFERENCES:
- [Background] Lindor KD, Gershwin ME, Poupon R, Kaplan M, Bergasa NV, Heathcote EJ; American Association for Study of Liver Diseases. Primary biliary cirrhosis. Hepatology. 2009 Jul;50(1):291-308. doi: 10.1002/hep.22906. No abstract available. PMID 19554543
- [Background] European Association for the Study of the Liver. EASL Clinical Practice Guidelines: management of cholestatic liver diseases. J Hepatol. 2009 Aug;51(2):237-67. doi: 10.1016/j.jhep.2009.04.009. Epub 2009 Jun 6. No abstract available. PMID 19501929
- [Background] Vilstrup H, Amodio P, Bajaj J, Cordoba J, Ferenci P, Mullen KD, Weissenborn K, Wong P. Hepatic encephalopathy in chronic liver disease: 2014 Practice Guideline by the American Association for the Study of Liver Diseases and the European Association for the Study of the Liver. Hepatology. 2014 Aug;60(2):715-35. doi: 10.1002/hep.27210. Epub 2014 Jul 8. No abstract available. PMID 25042402

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at study sites in the United States, Argentina, Belgium, Spain, Lithuania, Brazil, Australia, Germany, Estonia, Italy, Hungary, and Canada.
Pre-assignment Details: A total of 31 participants were screened and 22 participants were randomized.
Groups:
- Placebo: Participants received obeticholic acid (OCA) matching placebo tablets orally once weekly or twice weekly for the duration of at least 48 weeks. Participants, who had completed their 48-week treatment, could continue the treatment until all randomized participants had completed their 48-week treatment period and the database for that period was locked (total duration: approximately up to 3 years).
- Obeticholic Acid (OCA): Participants initiated treatment with OCA 5 milligrams (mg) tablets orally once weekly. At Week 12, if there were no safety concerns, the dose was up-titrated to OCA 5 mg twice weekly. Every 6 weeks thereafter, based on tolerability assessments, further up-titration of dose was considered. At each titration visit, the participants started the higher dose regimen no earlier than 2 days after the prior dose. The maximum dose titration was OCA 10 mg twice weekly at least 3 days apart. The minimum treatment duration was 48 weeks. Participants, who had completed their 48-week treatment, could continue the treatment until all randomized participants had completed their 48-week treatment period and the database for that period was locked (total duration: approximately up to 3 years).
Period: Double Blind (DB), up to Week 48
Arm/Group | Placebo | Obeticholic Acid (OCA)
Started | 12 | 10
Completed | 4 | 6
Not Completed | 8 | 4
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Death | 2 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Study Terminated by Sponsor | 2 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Liver Transplant During the Course of the Study | 1 | 0
Not completed — Multiple Serious Adverse Events and Drug Interruptions | 1 | 0
Period: DB Extension, Week 48 up to 3 Years
Arm/Group | Placebo | Obeticholic Acid (OCA)
Started | 4 | 6
Completed | 0 | 0
Not Completed | 4 | 6
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Death | 0 | 1
Not completed — Study Terminated by Sponsor | 3 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Intent-to-treat (ITT) population included all randomized participants who received any amount of investigational product (OCA or placebo).
Groups:
- Placebo: Participants received OCA matching placebo tablets orally once weekly or twice weekly for the duration of at least 48-weeks. Participants, who had completed their 48-week treatment, could continue the treatment until all randomized participants had completed their 48-week treatment period and the database for that period was locked (total duration: approximately up to 3 years).
- Obeticholic Acid (OCA): Participants initiated treatment with OCA 5 mg tablets orally once weekly. At Week 12, if there were no safety concerns, the dose was up-titrated to OCA 5 mg twice weekly. Every 6 weeks thereafter, based on tolerability assessments, further up-titration of dose was considered. At each titration visit, the participants started the higher dose regimen no earlier than 2 days after the prior dose. The maximum dose titration was OCA 10 mg twice weekly at least 3 days apart. The minimum treatment duration was 48-weeks. Participants, who had completed their 48-week treatment, could continue the treatment until all randomized participants had completed their 48-week treatment period and the database for that period was locked (total duration: approximately up to 3 years).
- Total: Total of all reporting groups
Arm/Group | Placebo | Obeticholic Acid (OCA) | Total
Number analyzed (Participants) | 12 | 10 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (9.10) | 60.5 (10.19) | 61.6 (9.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 16
  Male | 2 | 4 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 10
  Not Hispanic or Latino | 6 | 6 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 10 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Concentration (Cmax) of Total OCA at Week 12
Description: Total OCA is molar sum of unconjugated OCA, glyco-OCA, and tauro-OCA. Pharmacokinetics (PK) of OCA 5 mg twice weekly or 10 mg twice weekly at Week 12 are not applicable as no participant started 5 mg twice weekly or 10 mg twice weekly at Week 12.
Time Frame: Pre-dose (30 minutes before administration) and 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 9, and 24 hours post-dose at Week 12
Population: PK Population: participants who received OCA and had adequate concentration-time profile to characterize OCA and its conjugates and must not have had any major protocol deviations that potentially affect exposure level. Results of PK were planned to be listed by dose regimen. Participants who received planned dose regimen and had available data were included in the analysis. No participant started OCA 5 mg twice weekly or 10 mg twice weekly at Week 12.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Groups:
- OCA 5 mg Once Weekly: Participants received OCA 5 mg tablets orally once weekly.
- OCA 5 mg Twice Weekly: Participants received OCA 5 mg tablets orally twice weekly.
- OCA 10 mg Twice Weekly: Participants received OCA 10 mg tablets orally twice weekly.
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 5 | 0 | 0
nanogram per milliliter (ng/mL) | 293 (189) |  |

2. Primary Outcome: Time to Maximum Concentration (Tmax) of Total OCA at Week 12
Description: Total OCA is molar sum of unconjugated OCA, glyco-OCA, and tauro-OCA.
Time Frame: as for outcome 1
Population: Results of PK were planned to be listed by the dose regimen. Participants in the PK population who received the planned dose regimen and had available data were included in the analysis. Pharmacokinetics of OCA 5 mg twice weekly or 10 mg twice weekly at Week 12 are not applicable as no participant started 5 mg twice weekly or 10 mg twice weekly at Week 12.
Measure: Median (Full Range); unit: hours
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 5 | 0 | 0
hours | 2.02 [2.00 to 3.00] |  |

3. Primary Outcome: Trough Concentration (Ctrough) of Total OCA at Week 12
Description: Ctrough was considered as the concentration at 24-hours post-dose at Week 12. Total OCA is molar sum of unconjugated OCA, glyco-OCA, and tauro-OCA.
Time Frame: 24 hours post-dose at Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 4 | 0 | 0
ng/mL | 77.6 (49.7) |  |

4. Primary Outcome: Area Under the Concentration Versus Time Curve From Zero Time to 24 Hours (AUC0-24h) of Total OCA at Week 12
Description: Total OCA is molar sum of unconjugated OCA, glyco-OCA, and tauro-OCA. AUC0-24h was calculated using the linear/linear trapezoidal rule.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 4 | 0 | 0
nanogram*hour per milliliter (ng*h/mL) | 2970 (1650) |  |

5. Primary Outcome: Cmax of Total OCA at Week 18
Description: Total OCA is molar sum of unconjugated OCA, glyco-OCA, and tauro-OCA.
Time Frame: Pre-dose (30 minutes before administration) and 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 9, and 24 hours post-dose at Week 18
Population: Results of PK were planned to be listed by the dose regimen. Participants in the PK population who received the planned dose regimen and had available data were included in the analysis. Pharmacokinetics of OCA 10 mg twice weekly at Week 18 is not applicable as no participant started 10 mg twice weekly at Week 18.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 2 | 2 | 0
ng/mL | 136 (77.6) | 406 (120) |

6. Primary Outcome: Tmax of Total OCA at Week 18
Description: Total OCA is molar sum of unconjugated OCA, glyco-OCA, and tauro-OCA.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Median (Full Range); unit: hours
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 2 | 2 | 0
hours | 0.750 [0.500 to 1.00] | 2.52 [2.00 to 3.03] |

7. Primary Outcome: Ctrough of Total OCA at Week 18
Description: Ctrough was considered as the concentration at 24-hours post-dose at Week 18. Total OCA is molar sum of unconjugated OCA, glyco-OCA, and tauro-OCA.
Time Frame: 24 hours post-dose at Week 18
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 2 | 2 | 0
ng/mL | 28.7 (13.6) | 187 (147) |

8. Primary Outcome: AUC0-24h of Total OCA at Week 18
Description: as for outcome 4
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 2 | 2 | 0
ng*h/mL | 1380 (776) | 5810 (3600) |

9. Primary Outcome: Cmax of Total OCA at Week 24
Description: Total OCA is molar sum of unconjugated OCA, glyco-OCA, and tauro-OCA.
Time Frame: Pre-dose (30 minutes before administration) and 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 9, and 24 hours post-dose at Week 24
Population: Results of PK were planned to be listed by the dose regimen. Participants in the PK population who received the planned dose regimen and had available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 2 | 1 | 2
ng/mL | 263 (261) | 195 | 622 (117)

10. Primary Outcome: Tmax of Total OCA at Week 24
Description: Total OCA is molar sum of unconjugated OCA, glyco-OCA, and tauro-OCA.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Median (Full Range); unit: hours
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 2 | 1 | 2
hours | 5.04 [4.00 to 6.08] | 0.750 [0.750 to 0.750] | 2.27 [2.00 to 2.53]

11. Primary Outcome: Ctrough of Total OCA at Week 24
Description: Ctrough was considered as the concentration at 24-hours post-dose at Week 24. Total OCA is molar sum of unconjugated OCA, glyco-OCA, and tauro-OCA.
Time Frame: 24 hours post-dose at Week 24
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 2 | 1 | 2
ng/mL | 132 (163) | 41.4 | 435 (28.6)

12. Primary Outcome: AUC0-24h of Total OCA at Week 24
Description: as for outcome 4
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 2 | 1 | 2
ng*h/mL | 4500 (4910) | 2020 | 11300 (2950)

13. Primary Outcome: Cmax of Total OCA at Week 30
Description: Total OCA is molar sum of unconjugated OCA, glyco-OCA, and tauro-OCA.
Time Frame: Pre-dose (30 minutes before administration) and 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 9, and 24 hours post-dose at Week 30
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 1 | 2 | 2
ng/mL | 125 | 277 (64.7) | 674 (310)

14. Primary Outcome: Tmax of Total OCA at Week 30
Description: Total OCA is molar sum of unconjugated OCA, glyco-OCA, and tauro-OCA.
Time Frame: as for outcome 13
Population: as for outcome 9
Measure: Median (Full Range); unit: hours
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 1 | 2 | 2
hours | 1.00 [1.00 to 1.00] | 4.52 [4.03 to 5.00] | 3.77 [2.53 to 5.00]

15. Primary Outcome: Ctrough of Total OCA at Week 30
Description: Ctrough was considered as the concentration at 24-hours post-dose at Week 30. Total OCA is molar sum of unconjugated OCA, glyco-OCA, and tauro-OCA.
Time Frame: 24 hours post-dose at Week 30
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 1 | 2 | 2
ng/mL | 22.3 | 217 (15.7) | 317 (248)

16. Primary Outcome: AUC0-24h of Total OCA at Week 30
Description: as for outcome 4
Time Frame: as for outcome 13
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 1 | 2 | 2
ng*h/mL | 1260 | 5040 (855) | 10500 (7000)

17. Primary Outcome: Cmax of Total OCA at Week 48
Description: Total OCA is molar sum of unconjugated OCA, glyco-OCA, and tauro-OCA.
Time Frame: Pre-dose (30 minutes before administration) and 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 9, and 24 hours post-dose at Week 48
Population: Results of PK were planned to be listed by the dose regimen. Participants in the PK population who received the planned dose regimen and had available data were included in the analysis. Pharmacokinetics of OCA 5 mg once weekly at Week 48 is not applicable as participants received either OCA 5 mg twice daily or 10 mg twice daily and no participant received OCA 5 mg once weekly at Week 48.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 0 | 2 | 2
ng/mL |  | 200 (15.1) | 728 (27.5)

18. Primary Outcome: Tmax of Total OCA at Week 48
Description: Total OCA is molar sum of unconjugated OCA, glyco-OCA, and tauro-OCA.
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Median (Full Range); unit: hours
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 0 | 2 | 2
hours |  | 1.73 [1.47 to 2.00] | 4.03 [2.00 to 6.05]

19. Primary Outcome: Ctrough of Total OCA at Week 48
Description: Ctrough was considered as the concentration at 24-hours post-dose at Week 48. Total OCA is molar sum of unconjugated OCA, glyco-OCA, and tauro-OCA.
Time Frame: 24 hours post-dose at Week 48
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 0 | 2 | 2
ng/mL |  | 88.3 (29.9) | 497 (135)

20. Primary Outcome: AUC0-24h of Total OCA at Week 48
Description: as for outcome 4
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 0 | 2 | 2
ng*h/mL |  | 3210 (56.7) | 13900 (452)

21. Primary Outcome: Cmax of Unconjugated OCA at Week 12
Time Frame: as for outcome 1
Population: Results of PK were planned to be listed by dose regimen. Participants who received planned dose regimen and had available data were included in the analysis. Pharmacokinetics of OCA 5 mg twice weekly or 10 mg twice weekly at Week 12 are not applicable as no participant started 5 mg twice weekly or 10 mg twice weekly at Week 12.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 5 | 0 | 0
ng/mL | 107 (62.0) |  |

22. Primary Outcome: Tmax of Unconjugated OCA at Week 12
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 5 | 0 | 0
hours | 1.43 [1.00 to 1.50] |  |

23. Primary Outcome: Ctrough of Unconjugated OCA at Week 12
Description: Ctrough was considered as the concentration at 24-hours post-dose at Week 12.
Time Frame: 24 hours post-dose at Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 4 | 0 | 0
ng/mL | 2.92 (2.51) |  |

24. Primary Outcome: AUC0-24h of Unconjugated OCA at Week 12
Description: AUC0-24 was calculated using the linear/linear trapezoidal rule.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 3 | 0 | 0
ng*h/mL | 278 (142) |  |

25. Primary Outcome: Cmax of Unconjugated OCA at Week 18
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 2 | 2 | 0
ng/mL | 107 (47.4) | 109 (90.3) |

26. Primary Outcome: Tmax of Unconjugated OCA at Week 18
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Median (Full Range); unit: hours
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 2 | 2 | 0
hours | 0.750 [0.500 to 1.00] | 1.24 [1.00 to 1.48] |

27. Primary Outcome: Ctrough of Unconjugated OCA at Week 18
Description: Ctrough was considered as the concentration at 24-hours post-dose at Week 18.
Time Frame: 24 hours post-dose at Week 18
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 2 | 2 | 0
ng/mL | 3.38 (0.262) | 3.56 (4.01) |

28. Primary Outcome: AUC0-24h of Unconjugated OCA at Week 18
Description: AUC0-24h was calculated using the linear/linear trapezoidal rule.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 2 | 2 | 0
ng*h/mL | 191 (125) | 263 (247) |

29. Primary Outcome: Cmax of Unconjugated OCA at Week 24
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 2 | 1 | 2
ng/mL | 115 (98.2) | 157 | 168 (92.6)

30. Primary Outcome: Tmax of Unconjugated OCA at Week 24
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Median (Full Range); unit: hours
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 2 | 1 | 2
hours | 1.13 [0.750 to 1.50] | 0.500 [0.500 to 0.500] | 1.63 [1.58 to 1.67]

31. Primary Outcome: Ctrough of Unconjugated OCA at Week 24
Description: Ctrough was considered as the concentration at 24-hours post-dose at Week 24.
Time Frame: 24 hours post-dose at Week 24
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 2 | 1 | 2
ng/mL | 2.46 (2.05) | 5.18 | 8.77 (11.4)

32. Primary Outcome: AUC0-24h of Unconjugated OCA at Week 24
Description: AUC0-24h was calculated using the linear/linear trapezoidal rule.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 2 | 1 | 2
ng*h/mL | 235 (130) | 345 | 480 (414)

33. Primary Outcome: Cmax of Unconjugated OCA at Week 30
Time Frame: as for outcome 13
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 1 | 2 | 2
ng/mL | 92.6 | 132 (24.0) | 115 (40.9)

34. Primary Outcome: Tmax of Unconjugated OCA at Week 30
Time Frame: as for outcome 13
Population: as for outcome 9
Measure: Median (Full Range); unit: hours
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 1 | 2 | 2
hours | 0.750 [0.750 to 0.750] | 1.17 [1.00 to 1.33] | 1.75 [0.500 to 3.00]

35. Primary Outcome: Ctrough of Unconjugated OCA at Week 30
Description: Ctrough was considered as the concentration at 24-hours post-dose at Week 30.
Time Frame: 24 hours post-dose at Week 30
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 1 | 2 | 2
ng/mL | 3.03 | 4.27 (4.85) | 3.20 (3.14)

36. Primary Outcome: AUC0-24h of Unconjugated OCA at Week 30
Description: AUC0-24h was calculated using the linear/linear trapezoidal rule.
Time Frame: as for outcome 13
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 1 | 2 | 2
ng*h/mL | 176 | 304 (82.3) | 473 (397)

37. Primary Outcome: Cmax of Unconjugated OCA at Week 48
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 0 | 2 | 2
ng/mL |  | 131 (31.8) | 284 (177)

38. Primary Outcome: Tmax of Unconjugated OCA at Week 48
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Median (Full Range); unit: hours
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 0 | 2 | 2
hours |  | 1.10 [0.700 to 1.50] | 0.500 [0.500 to 0.500]

39. Primary Outcome: Ctrough of Unconjugated OCA at Week 48
Description: Ctrough was considered as the concentration at 24-hours post-dose at Week 48.
Time Frame: 24 hours post-dose at Week 48
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 0 | 2 | 2
ng/mL |  | 3.43 (3.90) | 4.72 (6.67)

40. Primary Outcome: AUC0-24h of Unconjugated OCA at Week 48
Description: AUC0-24h was calculated using the linear/linear trapezoidal rule.
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 0 | 2 | 1
ng*h/mL |  | 376 (118) | 1190

41. Primary Outcome: Cmax of Glyco Conjugate of OCA (Glyco-OCA) at Week 12
Time Frame: as for outcome 1
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 5 | 0 | 0
ng/mL | 117 (55.0) |  |

42. Primary Outcome: Tmax of Glyco-OCA at Week 12
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 5 | 0 | 0
hours | 5.00 [3.92 to 5.00] |  |

43. Primary Outcome: Ctrough of Glyco-OCA at Week 12
Description: Ctrough was considered as the concentration at 24-hours post-dose at Week 12.
Time Frame: 24 hours post-dose at Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 4 | 0 | 0
ng/mL | 47.1 (31.1) |  |

44. Primary Outcome: AUC0-24h of Glyco-OCA at Week 12
Description: AUC0-24h was calculated using the linear/linear trapezoidal rule.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 4 | 0 | 0
ng*h/mL | 1690 (947) |  |

45. Primary Outcome: Metabolite to Parent Ratio of AUC-0-24h (MRAUC) of Glyco-OCA at Week 12
Description: MRAUC was the ratio of AUC0-24h of Glyco-OCA (metabolite) to AUC0-24h of OCA (parent drug) * ratio of molecular weight of OCA to molecular weight of Glyco-OCA, where AUC0-24 is the area under the plasma concentration time profile from time 0 to 24 hours.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 3 | 0 | 0
ratio | 4.36 (1.03) |  |

46. Primary Outcome: Metabolite to Parent Ratio of Cmax (MRCmax) of Glyco-OCA at Week 12
Description: MRCmax was the ratio of Cmax of Glyco-OCA (metabolite) to Cmax of OCA (parent drug) * ratio of molecular weight of OCA to molecular weight of Glyco-OCA, where Cmax is the maximum observed concentration.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 5 | 0 | 0
ratio | 1.39 (1.38) |  |

47. Primary Outcome: Cmax of Glyco-OCA at Week 18
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 2 | 2 | 0
ng/mL | 52.7 (4.31) | 213 (22.6) |

48. Primary Outcome: Tmax of Glyco-OCA at Week 18
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Median (Full Range); unit: hours
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 2 | 2 | 0
hours | 4.25 [2.50 to 6.00] | 2.52 [2.00 to 3.03] |

49. Primary Outcome: Ctrough of Glyco-OCA at Week 18
Description: Ctrough was considered as the concentration at 24-hours post-dose at Week 18.
Time Frame: 24 hours post-dose at Week 18
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 2 | 2 | 0
ng/mL | 13.3 (5.03) | 98.1 (53.7) |

50. Primary Outcome: AUC0-24h of Glyco-OCA at Week 18
Description: AUC0-24h was calculated using the linear/linear trapezoidal rule.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 2 | 2 | 0
ng*h/mL | 625 (147) | 3020 (1120) |

51. Primary Outcome: MRAUC of Glyco-OCA at Week 18
Description: as for outcome 45
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 2 | 2 | 0
ratio | 3.39 (1.55) | 21.2 (23.6) |

52. Primary Outcome: MRCmax of Glyco-OCA at Week 18
Description: as for outcome 46
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 2 | 2 | 0
ratio | 0.487 (0.250) | 2.73 (2.44) |

53. Primary Outcome: Cmax of Glyco-OCA at Week 24
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 2 | 1 | 2
ng/mL | 166 (163) | 56.2 | 294 (70.0)

54. Primary Outcome: Tmax of Glyco-OCA at Week 24
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Median (Full Range); unit: hours
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 2 | 1 | 2
hours | 5.04 [4.00 to 6.08] | 5.00 [5.00 to 5.00] | 4.54 [4.08 to 5.00]

55. Primary Outcome: Ctrough of Glyco-OCA at Week 24
Description: Ctrough was considered as the concentration at 24-hours post-dose at Week 24.
Time Frame: 24 hours post-dose at Week 24
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 2 | 1 | 2
ng/mL | 83.0 (106) | 22.0 | 239 (7.07)

56. Primary Outcome: AUC0-24h of Glyco-OCA at Week 24
Description: AUC0-24h was calculated using the linear/linear trapezoidal rule.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 2 | 1 | 2
ng*h/mL | 2710 (3030) | 936 | 5550 (878)

57. Primary Outcome: MRAUC of Glyco-OCA at Week 24
Description: as for outcome 45
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 2 | 1 | 2
ratio | 8.26 (6.80) | 2.39 | 17.3 (16.5)

58. Primary Outcome: MRCmax of Glyco-OCA at Week 24
Description: as for outcome 46
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 2 | 1 | 2
ratio | 1.17 (0.253) | 0.315 | 1.94 (1.44)

59. Primary Outcome: Cmax of Glyco-OCA at Week 30
Time Frame: as for outcome 13
Population: Results of PK were planned to be listed by dose regimen. Participants who received planned dose regimen and had available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 1 | 2 | 2
ng/mL | 83.0 | 174 (75.0) | 301 (86.3)

60. Primary Outcome: Tmax of Glyco-OCA at Week 30
Time Frame: as for outcome 13
Population: as for outcome 9
Measure: Median (Full Range); unit: hours
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 1 | 2 | 2
hours | 6.00 [6.00 to 6.00] | 14.0 [4.03 to 24.0] | 4.51 [4.02 to 5.00]

61. Primary Outcome: Ctrough of Glyco-OCA at Week 30
Description: Ctrough was considered as the concentration at 24-hours post-dose at Week 30.
Time Frame: 24 hours post-dose at Week 30
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 1 | 2 | 2
ng/mL | 14.4 | 143 (30.4) | 156 (79.4)

62. Primary Outcome: AUC0-24h of Glyco-OCA at Week 30
Description: AUC0-24h was calculated using the linear/linear trapezoidal rule.
Time Frame: as for outcome 13
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 1 | 2 | 2
ng*h/mL | 863 | 3180 (1080) | 5050 (2260)

63. Primary Outcome: MRAUC of Glyco-OCA at Week 30
Description: as for outcome 45
Time Frame: as for outcome 13
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 1 | 2 | 2
ratio | 4.31 | 10.0 (5.84) | 17.2 (18.7)

64. Primary Outcome: MRCmax of Glyco-OCA at Week 30
Description: as for outcome 46
Time Frame: as for outcome 13
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 1 | 2 | 2
ratio | 0.789 | 1.23 (0.723) | 2.58 (1.58)

65. Primary Outcome: Cmax of Glyco-OCA at Week 48
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 0 | 2 | 2
ng/mL |  | 123 (34.0) | 354 (37.5)

66. Primary Outcome: Tmax of Glyco-OCA at Week 48
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Median (Full Range); unit: hours
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 0 | 2 | 2
hours |  | 5.00 [5.00 to 5.00] | 4.03 [2.00 to 6.05]

67. Primary Outcome: Ctrough of Glyco-OCA at Week 48
Description: Ctrough was considered as the concentration at 24-hours post-dose at Week 48.
Time Frame: 24 hours post-dose at Week 48
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 0 | 2 | 2
ng/mL |  | 65.9 (10.2) | 280 (62.2)

68. Primary Outcome: AUC0-24h of Glyco-OCA at Week 48
Description: AUC0-24h was calculated using the linear/linear trapezoidal rule.
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 0 | 2 | 2
ng*h/mL |  | 2120 (422) | 6950 (648)

69. Primary Outcome: MRAUC of Glyco-OCA at Week 48
Description: as for outcome 45
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 0 | 2 | 1
ratio |  | 5.39 (2.69) | 4.79

70. Primary Outcome: MRCmax of Glyco-OCA at Week 48
Description: as for outcome 46
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 0 | 2 | 2
ratio |  | 0.826 (0.0280) | 1.41 (1.00)

71. Primary Outcome: Cmax of Tauro Conjugate of OCA (Tauro-OCA) at Week 12
Time Frame: as for outcome 1
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 5 | 0 | 0
ng/mL | 201 (213) |  |

72. Primary Outcome: Tmax of Tauro-OCA at Week 12
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 5 | 0 | 0
hours | 5.00 [3.00 to 5.00] |  |

73. Primary Outcome: Ctrough of Tauro-OCA at Week 12
Description: Ctrough was considered as the concentration at 24-hours post-dose at Week 12.
Time Frame: 24 hours post-dose at Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 4 | 0 | 0
ng/mL | 41.6 (33.0) |  |

74. Primary Outcome: AUC0-24h of Tauro-OCA at Week 12
Description: AUC0-24h was calculated using the linear/linear trapezoidal rule.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 4 | 0 | 0
ng*h/mL | 1580 (1260) |  |

75. Primary Outcome: MRAUC of Tauro-OCA at Week 12
Description: MRAUC was the ratio of AUC0-24h of Tauro-OCA (metabolite) to AUC0-24h of OCA (parent drug) * ratio of molecular weight of OCA to molecular weight of Tauro-OCA, where AUC0-24 is the area under the plasma concentration time profile from time 0 to 24 hours.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 3 | 0 | 0
ratio | 3.13 (1.08) |  |

76. Primary Outcome: MRCmax of Tauro-OCA at Week 12
Description: MRCmax was the ratio of Cmax of Tauro-OCA (metabolite) to Cmax of OCA (parent drug) * ratio of molecular weight of OCA to molecular weight of Tauro-OCA, where Cmax is the maximum observed concentration.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 5 | 0 | 0
ratio | 2.24 (2.46) |  |

77. Primary Outcome: Cmax of Tauro-OCA at Week 18
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 2 | 2 | 0
ng/mL | 63.2 (46.9) | 221 (188) |

78. Primary Outcome: Tmax of Tauro-OCA at Week 18
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Median (Full Range); unit: hours
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 2 | 2 | 0
hours | 5.00 [5.00 to 5.00] | 2.52 [2.00 to 3.03] |

79. Primary Outcome: Ctrough of Tauro-OCA at Week 18
Description: Ctrough was considered as the concentration at 24-hours post-dose at Week 18.
Time Frame: 24 hours post-dose at Week 18
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 2 | 2 | 0
ng/mL | 17.0 (11.2) | 122 (130) |

80. Primary Outcome: AUC0-24h of Tauro-OCA at Week 18
Description: AUC0-24h was calculated using the linear/linear trapezoidal rule.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 2 | 2 | 0
ng*h/mL | 799 (654) | 3630 (3600) |

81. Primary Outcome: MRAUC of Tauro-OCA at Week 18
Description: as for outcome 75
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 2 | 2 | 0
ratio | 3.11 (0.685) | 28.8 (37.9) |

82. Primary Outcome: MRCmax of Tauro-OCA at Week 18
Description: as for outcome 76
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 2 | 2 | 0
ratio | 0.434 (0.156) | 3.32 (4.12) |

83. Primary Outcome: Cmax of Tauro-OCA at Week 24
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 2 | 1 | 2
ng/mL | 142 (144) | 65.5 | 430 (142)

84. Primary Outcome: Tmax of Tauro-OCA at Week 24
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Median (Full Range); unit: hours
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 2 | 1 | 2
hours | 5.54 [5.00 to 6.08] | 9.00 [9.00 to 9.00] | 4.05 [3.10 to 5.00]

85. Primary Outcome: Ctrough of Tauro-OCA at Week 24
Description: Ctrough was considered as the concentration at 24-hours post-dose at Week 24.
Time Frame: 24 hours post-dose at Week 24
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 2 | 1 | 2
ng/mL | 71.0 (90.5) | 21.2 | 271 (58.0)

86. Primary Outcome: AUC0-24h of Tauro-OCA at Week 24
Description: AUC0-24h was calculated using the linear/linear trapezoidal rule.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 2 | 1 | 2
ng*h/mL | 2360 (2650) | 1060 | 7470 (3260)

87. Primary Outcome: MRAUC of Tauro-OCA at Week 24
Description: as for outcome 75
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 2 | 1 | 2
ratio | 6.51 (5.40) | 2.46 | 23.4 (25.6)

88. Primary Outcome: MRCmax of Tauro-OCA at Week 24
Description: as for outcome 76
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 2 | 1 | 2
ratio | 0.881 (0.249) | 0.332 | 2.63 (2.13)

89. Primary Outcome: Cmax of Tauro-OCA at Week 30
Time Frame: as for outcome 13
Population: as for outcome 59
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 1 | 2 | 2
ng/mL | 38.6 | 141 (13.4) | 460 (342)

90. Primary Outcome: Tmax of Tauro-OCA at Week 30
Time Frame: as for outcome 13
Population: as for outcome 9
Measure: Median (Full Range); unit: hours
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 1 | 2 | 2
hours | 6.00 [6.00 to 6.00] | 4.52 [4.03 to 5.00] | 4.03 [3.05 to 5.00]

91. Primary Outcome: Ctrough of Tauro-OCA at Week 30
Description: Ctrough was considered as the concentration at 24-hours post-dose at Week 30.
Time Frame: 24 hours post-dose at Week 30
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 1 | 2 | 2
ng/mL | 8.21 | 110 (7.78) | 222 (228)

92. Primary Outcome: AUC0-24h of Tauro-OCA at Week 30
Description: AUC0-24h was calculated using the linear/linear trapezoidal rule.
Time Frame: as for outcome 13
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 1 | 2 | 2
ng*h/mL | 408 | 2430 (18.1) | 7020 (6780)

93. Primary Outcome: MRAUC of Tauro-OCA at Week 30
Description: as for outcome 75
Time Frame: as for outcome 13
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 1 | 2 | 2
ratio | 1.84 | 6.61 (1.74) | 25.7 (33.0)

94. Primary Outcome: MRCmax of Tauro-OCA at Week 30
Description: as for outcome 76
Time Frame: as for outcome 13
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 1 | 2 | 2
ratio | 0.332 | 0.855 (0.0746) | 3.85 (3.73)

95. Primary Outcome: Cmax of Tauro-OCA at Week 48
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 0 | 2 | 2
ng/mL |  | 72.5 (15.1) | 485 (20.5)

96. Primary Outcome: Tmax of Tauro-OCA at Week 48
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Median (Full Range); unit: hours
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 0 | 2 | 2
hours |  | 6.50 [6.00 to 7.00] | 2.57 [2.00 to 3.13]

97. Primary Outcome: Ctrough of Tauro-OCA at Week 48
Description: Ctrough was considered as the concentration at 24-hours post-dose at Week 48.
Time Frame: 24 hours post-dose at Week 48
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 0 | 2 | 2
ng/mL |  | 33.7 (21.4) | 309 (109)

98. Primary Outcome: AUC0-24h of Tauro-OCA at Week 48
Description: AUC0-24h was calculated using the linear/linear trapezoidal rule.
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 0 | 2 | 2
ng*h/mL |  | 1220 (389) | 8890 (696)

99. Primary Outcome: MRAUC of Tauro-OCA at Week 48
Description: as for outcome 75
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 0 | 2 | 1
ratio |  | 2.59 (0.00903) | 5.60

100. Primary Outcome: MRCmax of Tauro-OCA at Week 48
Description: as for outcome 76
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 0 | 2 | 2
ratio |  | 0.468 (0.206) | 1.67 (0.989)

101. Primary Outcome: Cmax of Glucuronide Metabolite of OCA (OCA-glucuronide) at Week 12
Time Frame: as for outcome 1
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 5 | 0 | 0
ng/mL | 47.0 (24.7) |  |

102. Primary Outcome: Tmax of OCA-glucuronide at Week 12
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 5 | 0 | 0
hours | 2.50 [1.50 to 3.00] |  |

103. Primary Outcome: Ctrough of OCA-glucuronide at Week 12
Description: Ctrough was considered as the concentration at 24-hours post-dose at Week 12.
Time Frame: 24 hours post-dose at Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 4 | 0 | 0
ng/mL | 20.7 (15.4) |  |

104. Primary Outcome: AUC0-24h of OCA-glucuronide at Week 12
Description: AUC0-24h was calculated using the linear/linear trapezoidal rule.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 4 | 0 | 0
ng*h/mL | 593 (388) |  |

105. Primary Outcome: MRAUC of OCA-glucuronide at Week 12
Description: MRAUC was the ratio of AUC0-24h of OCA-glucuronide (metabolite) to AUC0-24h of OCA (parent drug) * ratio of molecular weight of OCA to molecular weight of OCA-glucuronide, where AUC0-24 is the area under the plasma concentration time profile from time 0 to 24 hours.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 3 | 0 | 0
ratio | 1.17 (0.638) |  |

106. Primary Outcome: MRCmax of OCA-glucuronide at Week 12
Description: MRCmax was the ratio of Cmax of OCA-glucuronide (metabolite) to Cmax of OCA (parent drug) * ratio of molecular weight of OCA to molecular weight of OCA-glucuronide, where Cmax is the maximum observed concentration.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 5 | 0 | 0
ratio | 0.384 (0.275) |  |

107. Primary Outcome: Cmax of OCA-glucuronide at Week 18
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 2 | 2 | 0
ng/mL | 39.2 (30.3) | 74.9 (38.4) |

108. Primary Outcome: Tmax of OCA-glucuronide at Week 18
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Median (Full Range); unit: hours
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 2 | 2 | 0
hours | 1.25 [1.00 to 1.50] | 2.73 [1.50 to 3.97] |

109. Primary Outcome: Ctrough of OCA-glucuronide at Week 18
Description: Ctrough was considered as the concentration at 24-hours post-dose at Week 18.
Time Frame: 24 hours post-dose at Week 18
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 2 | 2 | 0
ng/mL | 11.7 (7.55) | 40.9 (43.9) |

110. Primary Outcome: AUC0-24h of OCA-glucuronide at Week 18
Description: AUC0-24h was calculated using the linear/linear trapezoidal rule.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 2 | 2 | 0
ng*h/mL | 390 (278) | 1120 (989) |

111. Primary Outcome: MRAUC of OCA-glucuronide at Week 18
Description: as for outcome 105
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 2 | 2 | 0
ratio | 1.41 (0.101) | 7.58 (9.76) |

112. Primary Outcome: MRCmax of OCA-glucuronide at Week 18
Description: as for outcome 106
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 2 | 2 | 0
ratio | 0.236 (0.0942) | 0.891 (0.985) |

113. Primary Outcome: Cmax of OCA-glucuronide at Week 24
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 2 | 1 | 2
ng/mL | 20.2 (7.42) | 58.1 | 127 (71.0)

114. Primary Outcome: Tmax of OCA-glucuronide at Week 24
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Median (Full Range); unit: hours
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 2 | 1 | 2
hours | 2.54 [2.08 to 3.00] | 1.00 [1.00 to 1.00] | 2.27 [2.00 to 2.53]

115. Primary Outcome: Ctrough of OCA-glucuronide at Week 24
Description: Ctrough was considered as the concentration at 24-hours post-dose at Week 24.
Time Frame: 24 hours post-dose at Week 24
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 2 | 1 | 2
ng/mL | 11.6 (6.43) | 14.5 | 84.2 (81.7)

116. Primary Outcome: AUC0-24h of OCA-glucuronide at Week 24
Description: AUC0-24h was calculated using the linear/linear trapezoidal rule.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 2 | 1 | 2
ng*h/mL | 330 (191) | 602 | 2120 (1920)

117. Primary Outcome: MRAUC of OCA-glucuronide at Week 24
Description: as for outcome 105
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 2 | 1 | 2
ratio | 0.983 (0.0286) | 1.23 | 6.87 (8.74)

118. Primary Outcome: MRCmax of OCA-glucuronide at Week 24
Description: as for outcome 106
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 2 | 1 | 2
ratio | 0.165 (0.0959) | 0.261 | 0.727 (0.701)

119. Primary Outcome: Cmax of OCA-glucuronide at Week 30
Time Frame: as for outcome 13
Population: as for outcome 59
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 1 | 2 | 2
ng/mL | 13.7 | 51.9 (49.4) | 148 (117)

120. Primary Outcome: Tmax of OCA-glucuronide at Week 30
Time Frame: as for outcome 13
Population: as for outcome 9
Measure: Median (Full Range); unit: hours
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 1 | 2 | 2
hours | 1.50 [1.50 to 1.50] | 2.26 [1.50 to 3.02] | 4.51 [4.02 to 5.00]

121. Primary Outcome: Ctrough of OCA-glucuronide at Week 30
Description: Ctrough was considered as the concentration at 24-hours post-dose at Week 30.
Time Frame: 24 hours post-dose at Week 30
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 1 | 2 | 2
ng/mL | 5.57 | 19.7 (13.8) | 89.0 (107)

122. Primary Outcome: AUC0-24h of OCA-glucuronide at Week 30
Description: AUC0-24h was calculated using the linear/linear trapezoidal rule.
Time Frame: as for outcome 13
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 1 | 2 | 2
ng*h/mL | 170 | 641 (482) | 2200 (2100)

123. Primary Outcome: MRAUC of OCA-glucuronide at Week 30
Description: as for outcome 105
Time Frame: as for outcome 13
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 1 | 2 | 2
ratio | 0.680 | 1.39 (0.742) | 7.10 (9.09)

124. Primary Outcome: MRCmax of OCA-glucuronide at Week 30
Description: as for outcome 106
Time Frame: as for outcome 13
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 1 | 2 | 2
ratio | 0.104 | 0.257 (0.217) | 1.11 (1.11)

125. Primary Outcome: Cmax of OCA-glucuronide at Week 48
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 0 | 2 | 2
ng/mL |  | 66.0 (63.6) | 134 (71.3)

126. Primary Outcome: Tmax of OCA-glucuronide at Week 48
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Median (Full Range); unit: hours
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 0 | 2 | 2
hours |  | 1.73 [1.47 to 2.00] | 1.54 [1.50 to 1.58]

127. Primary Outcome: Ctrough of OCA-glucuronide at Week 48
Description: Ctrough was considered as the concentration at 24-hours post-dose at Week 48.
Time Frame: 24 hours post-dose at Week 48
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 0 | 2 | 2
ng/mL |  | 39.2 (35.7) | 89.2 (73.3)

128. Primary Outcome: AUC0-24h of OCA-glucuronide at Week 48
Description: AUC0-24h was calculated using the linear/linear trapezoidal rule.
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 0 | 2 | 2
ng*h/mL |  | 952 (833) | 2490 (1520)

129. Primary Outcome: MRAUC of OCA-glucuronide at Week 48
Description: as for outcome 105
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 0 | 2 | 1
ratio |  | 1.62 (1.05) | 0.833

130. Primary Outcome: MRCmax of OCA-glucuronide at Week 48
Description: as for outcome 106
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | OCA 5 mg Once Weekly | OCA 5 mg Twice Weekly | OCA 10 mg Twice Weekly
Number analyzed (Participants) | 0 | 2 | 2
ratio |  | 0.411 (0.444) | 0.482 (0.479)

131. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not related to the study drug.
  An SAE was any AE that results in death, was life-threatening, resulted in a persistent or significant disability/incapacity, resulted in in-patient hospitalization or prolonged an existing hospitalization, was a congenital anomaly/birth defect, or was an important medical event that could jeopardize the participant or could have required medical intervention to prevent one of the outcomes listed above.
  TEAE was defined as any AE if it met one or more of the following criteria: 1) An AE started on or after the first study drug dose and within 30 days after the last dose of study drug, 2) An AE occurred prior to the first study drug dose that worsens (increase in grade) after the first study drug dose.
Time Frame: Baseline up to approximately 3 years
Population: The Safety Population included all participants who received at least 1 dose of investigational product (OCA or placebo). Data were prespecified to be collected per randomization arm (OCA or placebo). Data at the separate dose levels are not available.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Obeticholic Acid (OCA)
Number analyzed (Participants) | 12 | 10
Participants
  Any TEAE | 12 | 10
  SAE | 9 | 7

132. Secondary Outcome: Change From Baseline in the Model of End-stage Liver Disease (MELD) Score at Weeks 3, 6, 12, 18, 24, 30, 36, 42, and 48; and Extension Months 3, 6, 9, 12, and 15
Description: The MELD scoring system is used to assess the severity of chronic liver disease. The MELD score is derived from the participant's serum total bilirubin, serum creatinine, and prothrombin international normalized ratio (INR): 3.78×log normal (ln) [total bilirubin (mg/deciliter [dL])] + 11.2×ln[INR] + 9.57×ln[serum creatinine (mg/dL)] + 6.43. The MELD score ranges from 6 to 40 with higher scores indicating more severe liver disease and a worse outcome.
Time Frame: Baseline, Weeks 3, 6, 12, 18, 24, 30, 36, 42, and 48; and Extension Months 3, 6, 9, 12, and 15
Population: Participants in the ITT population with available data were analyzed. Data were prespecified to be collected per randomization arm (OCA or placebo). Data at the separate dose levels are not available.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Placebo: Participants received OCA matching placebo tablets orally once weekly or twice weekly for the duration of at least 48 weeks. Participants, who had completed their 48-week treatment, could continue the treatment until all randomized participants had completed their 48-week treatment period and the database for that period was locked (total duration: approximately up to 3 years).
- Obeticholic Acid (OCA): Participants initiated treatment with OCA 5 mg tablets orally once weekly. At Week 12, if there were no safety concerns, the dose was up-titrated to OCA 5 mg twice weekly. Every 6 weeks thereafter, based on tolerability assessments, further up-titration of dose was considered. At each titration visit, the participants started the higher dose regimen no earlier than 2 days after the prior dose. The maximum dose titration was OCA 10 mg twice weekly at least 3 days apart. The minimum treatment duration was 48 weeks. Participants, who had completed their 48-week treatment, could continue the treatment until all randomized participants had completed their 48-week treatment period and the database for that period was locked (total duration: approximately up to 3 years).
Arm/Group | Placebo | Obeticholic Acid (OCA)
Number analyzed (Participants) | 12 | 10
score on a scale
  Baseline | 11.75 [10.60 to 13.50] | 12.75 [9.50 to 16.00]
  Change at Week 3: number analyzed (Participants) | 11 | 10
  Change at Week 3 | 0.50 [-0.50 to 1.00] | 0.00 [-1.50 to 2.00]
  Change at Week 6: number analyzed (Participants) | 9 | 8
  Change at Week 6 | 0.50 [0.00 to 2.50] | 0.00 [-0.75 to 1.25]
  Change at Week 12: number analyzed (Participants) | 6 | 7
  Change at Week 12 | 0.75 [0.00 to 2.50] | 0.00 [-1.00 to 1.00]
  Change at Week 18: number analyzed (Participants) | 8 | 8
  Change at Week 18 | 0.65 [-0.25 to 3.00] | -0.75 [-2.00 to 1.00]
  Change at Week 24: number analyzed (Participants) | 4 | 5
  Change at Week 24 | 0.15 [0.00 to 0.40] | -1.50 [-2.00 to 0.00]
  Change at Week 30: number analyzed (Participants) | 6 | 6
  Change at Week 30 | 0.15 [-0.50 to 0.50] | -1.25 [-2.00 to 0.00]
  Change at Week 36: number analyzed (Participants) | 6 | 6
  Change at Week 36 | 0.15 [-1.00 to 1.50] | 0.25 [-1.50 to 1.00]
  Change at Week 42: number analyzed (Participants) | 6 | 6
  Change at Week 42 | 0.65 [-0.50 to 1.50] | 0.50 [0.00 to 1.50]
  Change at Week 48: number analyzed (Participants) | 6 | 4
  Change at Week 48 | 0.65 [0.00 to 1.50] | -1.75 [-2.50 to -0.50]
  Change at Extension Month 3: number analyzed (Participants) | 5 | 5
  Change at Extension Month 3 | 0.50 [0.50 to 4.30] | -1.00 [-1.50 to -0.50]
  Change at Extension Month 6: number analyzed (Participants) | 3 | 2
  Change at Extension Month 6 | 0.00 [-1.00 to 3.50] | 0.25 [0.00 to 0.50]
  Change at Extension Month 9: number analyzed (Participants) | 0 | 2
  Change at Extension Month 9 |  | 0.75 [-1.00 to 2.50]
  Change at Extension Month 12: number analyzed (Participants) | 1 | 1
  Change at Extension Month 12 | -1.00 [-1.00 to -1.00] | 4.50 [4.50 to 4.50]
  Change at Extension Month 15: number analyzed (Participants) | 1 | 0
  Change at Extension Month 15 | -1.00 [-1.00 to -1.00] |

133. Secondary Outcome: Change From Baseline in MELD-Sodium (Na) Score at Weeks 3, 6, 12, 18, 24, 30, 36, 42, and 48; and Extension Months 3, 6, 9, 12, and 15
Description: The MELD-Na scoring system is used to assess the severity of chronic liver disease in the participants with an initial MELD(i) score greater than 11. MELD-Na score is derived from the participant's serum total bilirubin, serum creatinine, INR, and sodium. The MELD-Na score is re-calculated as follows:
  MELD-Na = MELD(i) + 1.32*(137-Na) - [0.033*MELD(i)*(137-Na)]. MELD score ranges from 6-40 with higher scores indicating more severe liver disease and a worse outcome.
  The MELD(i) score is derived from the participant's serum total bilirubin, serum creatinine, and prothrombin international normalized ratio (INR): 3.78×log normal (ln) [total bilirubin (mg/deciliter [dL])] + 11.2×ln[INR] + 9.57×ln[serum creatinine (mg/dL)] + 6.43. The MELD score ranges from 6 to 40 with higher scores indicating more severe liver disease and a worse outcome.
Time Frame: Baseline, Weeks 3, 6, 12, 18, 24, 30, 36, 42, and 48; and Extension Months 3, 6, 9, 12, and 15
Population: as for outcome 132
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Placebo | Obeticholic Acid (OCA)
Number analyzed (Participants) | 12 | 10
score on a scale
  Baseline | 11.75 [10.60 to 14.25] | 13.25 [9.50 to 16.00]
  Change at Week 3: number analyzed (Participants) | 11 | 10
  Change at Week 3 | 0.00 [-0.50 to 1.00] | 0.50 [-1.50 to 2.00]
  Change at Week 6: number analyzed (Participants) | 9 | 8
  Change at Week 6 | 0.50 [0.00 to 2.00] | -0.25 [-0.75 to 1.50]
  Change at Week 12: number analyzed (Participants) | 6 | 7
  Change at Week 12 | 0.50 [0.00 to 3.50] | 0.50 [-1.50 to 2.00]
  Change at Week 18: number analyzed (Participants) | 8 | 8
  Change at Week 18 | 0.65 [-0.25 to 2.75] | -0.75 [-2.50 to 0.50]
  Change at Week 24: number analyzed (Participants) | 4 | 5
  Change at Week 24 | 0.15 [0.00 to 0.40] | -2.00 [-2.50 to 1.00]
  Change at Week 30: number analyzed (Participants) | 6 | 6
  Change at Week 30 | 0.15 [-0.50 to 0.50] | -0.75 [-2.00 to 0.50]
  Change at Week 36: number analyzed (Participants) | 6 | 6
  Change at Week 36 | 0.15 [-1.00 to 1.50] | -0.25 [-1.50 to 1.00]
  Change at Week 42: number analyzed (Participants) | 5 | 6
  Change at Week 42 | 0.00 [-0.50 to 1.30] | 0.50 [0.00 to 0.50]
  Change at Week 48: number analyzed (Participants) | 6 | 4
  Change at Week 48 | 0.65 [0.00 to 2.50] | -1.75 [-3.00 to 0.00]
  Change at Extension Month 3: number analyzed (Participants) | 5 | 5
  Change at Extension Month 3 | 2.50 [0.50 to 4.30] | -1.00 [-2.50 to -0.50]
  Change at Extension Month 6: number analyzed (Participants) | 3 | 2
  Change at Extension Month 6 | 0.00 [-1.00 to 3.50] | 1.75 [0.50 to 3.00]
  Change at Extension Month 9: number analyzed (Participants) | 0 | 2
  Change at Extension Month 9 |  | 0.75 [-1.00 to 2.50]
  Change at Extension Month 12: number analyzed (Participants) | 1 | 1
  Change at Extension Month 12 | -1.00 [-1.00 to -1.00] | 4.50 [4.50 to 4.50]
  Change at Extension Month 15: number analyzed (Participants) | 1 | 0
  Change at Extension Month 15 | -1.00 [-1.00 to -1.00] |

134. Secondary Outcome: Change From Baseline in Child-Pugh Score at Day 1, Weeks 6, 12, 18, 24, 30, 36, and 48; and Extension Months 3, 6, 9, 12, and 15
Description: The Child-Pugh classification was a scoring system used for the classification of the severity of cirrhosis. It included three continuous variables (bilirubin, albumin, and INR) and two discrete variables (ascites and encephalopathy). Each variable was scored 1-3 with 3 indicating most severe derangement. The determination of Child-Pugh score ranged from 5 to 15. The higher the score, the sicker the participant.
Time Frame: Baseline, Day 1, Weeks 6, 12, 18, 24, 30, 36, and 48; and Extension Months 3, 6, 9, 12, and 15
Population: as for outcome 132
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Placebo | Obeticholic Acid (OCA)
Number analyzed (Participants) | 12 | 10
score on a scale
  Baseline | 8.0 [7.0 to 8.0] | 8.0 [7.0 to 8.0]
  Change at Day 1 | 0.0 [-0.5 to 0.0] | 0.0 [0.0 to 0.0]
  Change at Week 6: number analyzed (Participants) | 9 | 8
  Change at Week 6 | 0.0 [-1.0 to 0.0] | 0.0 [-0.5 to 0.5]
  Change at Week 12: number analyzed (Participants) | 6 | 7
  Change at Week 12 | -0.5 [-1.0 to 1.0] | 0.0 [-1.0 to 1.0]
  Change at Week 18: number analyzed (Participants) | 8 | 8
  Change at Week 18 | 0.0 [-1.0 to 0.0] | -0.5 [-2.0 to 0.0]
  Change at Week 24: number analyzed (Participants) | 5 | 5
  Change at Week 24 | -1.0 [-1.0 to 0.0] | 0.0 [-1.0 to 0.0]
  Change at Week 30: number analyzed (Participants) | 6 | 6
  Change at Week 30 | -0.5 [-1.0 to 0.0] | -1.0 [-2.0 to 0.0]
  Change at Week 36: number analyzed (Participants) | 6 | 6
  Change at Week 36 | -1.0 [-1.0 to 0.0] | -0.5 [-1.0 to 0.0]
  Change at Week 48: number analyzed (Participants) | 6 | 6
  Change at Week 48 | -0.5 [-1.0 to 0.0] | 0.0 [-2.0 to 0.0]
  Change at Extension Month 3: number analyzed (Participants) | 6 | 5
  Change at Extension Month 3 | 0.0 [-1.0 to 0.0] | 0.0 [-1.0 to 1.0]
  Change at Extension Month 6: number analyzed (Participants) | 3 | 2
  Change at Extension Month 6 | 1.0 [-2.0 to 3.0] | 0.0 [0.0 to 0.0]
  Change at Extension Month 9: number analyzed (Participants) | 0 | 2
  Change at Extension Month 9 |  | 0.0 [-1.0 to 1.0]
  Change at Extension Month 12: number analyzed (Participants) | 1 | 1
  Change at Extension Month 12 | 1.0 [1.0 to 1.0] | 0.0 [0.0 to 0.0]
  Change at Extension Month 15: number analyzed (Participants) | 1 | 0
  Change at Extension Month 15 | 1.0 [1.0 to 1.0] |

135. Secondary Outcome: Number of Participants by Child-Pugh Score Component Category (Ascites Categories)
Description: Number of participants with Child-Pugh component - ascites categories of none, mild, and moderate-severe has been reported. The ascites categories were defined per investigator's discretion.
Time Frame: Day 1, Weeks 6, 12, 18, 24, 30, 36, and 48; and Extension Months 3, 6, 9, 12, and 15
Population: as for outcome 132
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Obeticholic Acid (OCA)
Number analyzed (Participants) | 12 | 10
Participants
  Baseline: None | 6 | 5
  Baseline: Mild | 5 | 3
  Baseline: Moderate-Severe | 1 | 2
  Day 1: None | 6 | 5
  Day 1: Mild | 5 | 4
  Day 1: Moderate-Severe | 1 | 1
  Week 6: number analyzed (Participants) | 9 | 9
  Week 6: None | 7 | 4
  Week 6: Mild | 2 | 5
  Week 6: Moderate-Severe | 0 | 0
  Week 12: number analyzed (Participants) | 6 | 7
  Week 12: None | 4 | 4
  Week 12: Mild | 2 | 3
  Week 12: Moderate-Severe | 0 | 0
  Week 18: number analyzed (Participants) | 8 | 8
  Week 18: None | 6 | 5
  Week 18: Mild | 2 | 3
  Week 18: Moderate-Severe | 0 | 0
  Week 24: number analyzed (Participants) | 6 | 6
  Week 24: None | 6 | 3
  Week 24: Mild | 0 | 3
  Week 24: Moderate-Severe | 0 | 0
  Week 30: number analyzed (Participants) | 6 | 6
  Week 30: None | 6 | 4
  Week 30: Mild | 0 | 2
  Week 30: Moderate-Severe | 0 | 0
  Week 36: number analyzed (Participants) | 6 | 6
  Week 36: None | 6 | 4
  Week 36: Mild | 0 | 2
  Week 36: Moderate-Severe | 0 | 0
  Week 48: number analyzed (Participants) | 6 | 6
  Week 48: None | 6 | 4
  Week 48: Mild | 0 | 1
  Week 48: Moderate-Severe | 0 | 1
  Extension Month 3: number analyzed (Participants) | 6 | 5
  Extension Month 3: None | 6 | 2
  Extension Month 3: Mild | 0 | 1
  Extension Month 3: Moderate-Severe | 0 | 2
  Extension Month 6: number analyzed (Participants) | 3 | 2
  Extension Month 6: None | 1 | 1
  Extension Month 6: Mild | 1 | 1
  Extension Month 6: Moderate-Severe | 1 | 0
  Extension Month 9: number analyzed (Participants) | 0 | 2
  Extension Month 9: None | 0 | 1
  Extension Month 9: Mild | 0 | 1
  Extension Month 9: Moderate-Severe | 0 | 0
  Extension Month 12: number analyzed (Participants) | 1 | 1
  Extension Month 12: None | 0 | 0
  Extension Month 12: Mild | 1 | 1
  Extension Month 12: Moderate-Severe | 0 | 0
  Extension Month 15: number analyzed (Participants) | 1 | 1
  Extension Month 15: None | 0 | 0
  Extension Month 15: Mild | 1 | 1
  Extension Month 15: Moderate-Severe | 0 | 0

136. Secondary Outcome: Number of Participants by Child-Pugh Score Component Category (Prothrombin Time Categories)
Description: Number of participants with Child-Pugh component - prothrombin time (measured as INR) in categories of <1.7, 1.7 - 2.3, and >2.3 has been reported.
Time Frame: Day 1, Weeks 6, 12, 18, 24, 30, 36, and 48; and Extension Months 3, 6, 9, 12, and 15
Population: as for outcome 132
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Obeticholic Acid (OCA)
Number analyzed (Participants) | 12 | 10
Participants
  Baseline: <1.7 | 12 | 10
  Baseline: 1.7 - 2.3 | 0 | 0
  Baseline: >2.3 | 0 | 0
  Day 1: <1.7 | 12 | 10
  Day 1: 1.7 - 2.3 | 0 | 0
  Day 1: >2.3 | 0 | 0
  Week 6: number analyzed (Participants) | 9 | 9
  Week 6: <1.7 | 9 | 9
  Week 6: 1.7 - 2.3 | 0 | 0
  Week 6: >2.3 | 0 | 0
  Week 12: number analyzed (Participants) | 6 | 7
  Week 12: <1.7 | 6 | 7
  Week 12: 1.7 - 2.3 | 0 | 0
  Week 12: >2.3 | 0 | 0
  Week 18: number analyzed (Participants) | 8 | 8
  Week 18: <1.7 | 8 | 8
  Week 18: 1.7 - 2.3 | 0 | 0
  Week 18: >2.3 | 0 | 0
  Week 24: number analyzed (Participants) | 5 | 5
  Week 24: <1.7 | 4 | 5
  Week 24: 1.7 - 2.3 | 1 | 0
  Week 24: >2.3 | 0 | 0
  Week 30: number analyzed (Participants) | 6 | 6
  Week 30: <1.7 | 6 | 6
  Week 30: 1.7 - 2.3 | 0 | 0
  Week 30: >2.3 | 0 | 0
  Week 36: number analyzed (Participants) | 6 | 6
  Week 36: <1.7 | 6 | 6
  Week 36: 1.7 - 2.3 | 0 | 0
  Week 36: >2.3 | 0 | 0
  Week 48: number analyzed (Participants) | 6 | 6
  Week 48: <1.7 | 6 | 6
  Week 48: 1.7 - 2.3 | 0 | 0
  Week 48: >2.3 | 0 | 0
  Extension Month 3: number analyzed (Participants) | 6 | 5
  Extension Month 3: <1.7 | 6 | 5
  Extension Month 3: 1.7 - 2.3 | 0 | 0
  Extension Month 3: >2.3 | 0 | 0
  Extension Month 6: number analyzed (Participants) | 3 | 2
  Extension Month 6: <1.7 | 3 | 2
  Extension Month 6: 1.7 - 2.3 | 0 | 0
  Extension Month 6: >2.3 | 0 | 0
  Extension Month 9: number analyzed (Participants) | 0 | 2
  Extension Month 9: <1.7 | 0 | 2
  Extension Month 9: 1.7 - 2.3 | 0 | 0
  Extension Month 9: >2.3 | 0 | 0
  Extension Month 12: number analyzed (Participants) | 1 | 1
  Extension Month 12: <1.7 | 1 | 1
  Extension Month 12: 1.7 - 2.3 | 0 | 0
  Extension Month 12: >2.3 | 0 | 0
  Extension Month 15: number analyzed (Participants) | 1 | 0
  Extension Month 15: <1.7 | 1 | 0
  Extension Month 15: 1.7 - 2.3 | 0 | 0
  Extension Month 15: >2.3 | 0 | 0

137. Secondary Outcome: Number of Participants by Child-Pugh Score Component Category (Serum Albumin Categories)
Description: Number of participants with Child-Pugh component - serum albumin levels in categories of >35 gram per liter (g/L), 28-35 g/L, or <28 g/L has been reported.
Time Frame: Day 1, Weeks 6, 12, 18, 24, 30, 36, and 48; and Extension Months 3, 6, 9, 12, and 15
Population: as for outcome 132
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Obeticholic Acid (OCA)
Number analyzed (Participants) | 12 | 10
Participants
  Baseline: >35 g/L | 3 | 4
  Baseline: 28 - 35 g/L | 8 | 5
  Baseline: <28 g/L | 1 | 1
  Day 1: >35 g/L | 3 | 4
  Day 1: 28 - 35 g/L | 9 | 4
  Day 1: <28 g/L | 0 | 2
  Week 12: number analyzed (Participants) | 6 | 7
  Week 12: >35 g/L | 1 | 3
  Week 12: 28 - 35 g/L | 5 | 3
  Week 12: <28 g/L | 0 | 1
  Week 6: number analyzed (Participants) | 9 | 9
  Week 6: >35 g/L | 2 | 4
  Week 6: 28 - 35 g/L | 7 | 3
  Week 6: <28 g/L | 0 | 2
  Week 18: number analyzed (Participants) | 8 | 8
  Week 18: >35 g/L | 2 | 5
  Week 18: 28 - 35 g/L | 6 | 3
  Week 18: <28 g/L | 0 | 0
  Week 24: number analyzed (Participants) | 6 | 6
  Week 24: >35 g/L | 1 | 3
  Week 24: 28 - 35 g/L | 5 | 3
  Week 24: <28 g/L | 0 | 0
  Week 30: number analyzed (Participants) | 6 | 6
  Week 30: >35 g/L | 1 | 3
  Week 30: 28 - 35 g/L | 5 | 3
  Week 30: <28 g/L | 0 | 0
  Week 36: number analyzed (Participants) | 6 | 6
  Week 36: >35 g/L | 1 | 2
  Week 36: 28 - 35 g/L | 5 | 4
  Week 36: <28 g/L | 0 | 0
  Week 48: number analyzed (Participants) | 6 | 6
  Week 48: >35 g/L | 2 | 3
  Week 48: 28 - 35 g/L | 4 | 3
  Week 48: <28 g/L | 0 | 0
  Extension Month 3: number analyzed (Participants) | 6 | 5
  Extension Month 3: >35 g/L | 1 | 2
  Extension Month 3: 28 - 35 g/L | 5 | 3
  Extension Month 3: <28 g/L | 0 | 0
  Extension Month 6: number analyzed (Participants) | 3 | 2
  Extension Month 6: >35 g/L | 1 | 1
  Extension Month 6: 28 - 35 g/L | 2 | 1
  Extension Month 6: <28 g/L | 0 | 0
  Extension Month 9: number analyzed (Participants) | 0 | 2
  Extension Month 9: >35 g/L | 0 | 0
  Extension Month 9: 28 - 35 g/L | 0 | 2
  Extension Month 9: <28 g/L | 0 | 0
  Extension Month 12: number analyzed (Participants) | 1 | 1
  Extension Month 12: >35 g/L | 0 | 1
  Extension Month 12: 28 - 35 g/L | 1 | 0
  Extension Month 12: <28 g/L | 0 | 0
  Extension Month 15: number analyzed (Participants) | 1 | 1
  Extension Month 15: >35 g/L | 0 | 0
  Extension Month 15: 28 - 35 g/L | 1 | 1
  Extension Month 15: <28 g/L | 0 | 0

138. Secondary Outcome: Number of Participants by Child-Pugh Score Component Category (Total Bilirubin Categories)
Description: Number of participants with Child-Pugh component - total bilirubin levels in categories of <34 micromole per liter (µmol/L), 34-50 µmol/L, and >50 µmol/L has been reported.
Time Frame: Day 1, Weeks 6, 12, 18, 24, 30, 36, and 48; and Extension Months 3, 6, 9, 12, and 15
Population: as for outcome 132
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Obeticholic Acid (OCA)
Number analyzed (Participants) | 12 | 10
Participants
  Baseline: <34 µmol/L | 3 | 5
  Baseline: 34-50 µmol/L | 5 | 0
  Baseline: >50 µmol/L | 4 | 5
  Day 1: <34 µmol/L | 3 | 5
  Day 1: 34-50 µmol/L | 5 | 0
  Day 1: >50 µmol/L | 4 | 5
  Week 6: number analyzed (Participants) | 9 | 8
  Week 6: <34 µmol/L | 4 | 4
  Week 6: 34-50 µmol/L | 1 | 0
  Week 6: >50 µmol/L | 4 | 4
  Week 12: number analyzed (Participants) | 6 | 7
  Week 12: <34 µmol/L | 2 | 4
  Week 12: 34-50 µmol/L | 3 | 0
  Week 12: >50 µmol/L | 1 | 3
  Week 18: number analyzed (Participants) | 8 | 8
  Week 18: <34 µmol/L | 2 | 5
  Week 18: 34-50 µmol/L | 3 | 0
  Week 18: >50 µmol/L | 3 | 3
  Week 24: number analyzed (Participants) | 6 | 6
  Week 24: <34 µmol/L | 2 | 4
  Week 24: 34-50 µmol/L | 3 | 0
  Week 24: >50 µmol/L | 1 | 2
  Week 30: number analyzed (Participants) | 6 | 6
  Week 30: <34 µmol/L | 3 | 4
  Week 30: 34-50 µmol/L | 1 | 1
  Week 30: >50 µmol/L | 2 | 1
  Week 36: number analyzed (Participants) | 6 | 6
  Week 36: <34 µmol/L | 3 | 4
  Week 36: 34-50 µmol/L | 1 | 0
  Week 36: >50 µmol/L | 2 | 2
  Week 48: number analyzed (Participants) | 6 | 6
  Week 48: <34 µmol/L | 2 | 4
  Week 48: 34-50 µmol/L | 1 | 0
  Week 48: >50 µmol/L | 3 | 2
  Extension Month 3: number analyzed (Participants) | 6 | 5
  Extension Month 3: <34 µmol/L | 2 | 3
  Extension Month 3: 34-50 µmol/L | 1 | 1
  Extension Month 3: >50 µmol/L | 3 | 1
  Extension Month 6: number analyzed (Participants) | 3 | 2
  Extension Month 6: <34 µmol/L | 1 | 1
  Extension Month 6: 34-50 µmol/L | 1 | 0
  Extension Month 6: >50 µmol/L | 1 | 1
  Extension Month 9: number analyzed (Participants) | 0 | 2
  Extension Month 9: <34 µmol/L | 0 | 1
  Extension Month 9: 34-50 µmol/L | 0 | 1
  Extension Month 9: >50 µmol/L | 0 | 0
  Extension Month 12: number analyzed (Participants) | 1 | 1
  Extension Month 12: <34 µmol/L | 0 | 1
  Extension Month 12: 34-50 µmol/L | 1 | 0
  Extension Month 12: >50 µmol/L | 0 | 0
  Extension Month 15: number analyzed (Participants) | 1 | 1
  Extension Month 15: <34 µmol/L | 0 | 1
  Extension Month 15: 34-50 µmol/L | 1 | 0
  Extension Month 15: >50 µmol/L | 0 | 0

139. Secondary Outcome: Number of Participants by Child-Pugh Score Component Category (Hepatic Encephalopathy Categories)
Description: Number of participants with Child-Pugh component - Hepatic encephalopathy in categories of Grade 0, Grade 1 or 2, and Grade 3 and 4 has been reported.
  Grade 0: normal consciousness, normal personality, normal neurological examination, normal electroencephalogram.
  Grade 1: restless, sleep disturbed, irritable/agitated, tremor, impaired handwriting, 5 cycles, per second (cps) waves.
  Grade 2: lethargic, time-disoriented, inappropriate, asterixis, ataxia, slow triphasic waves.
  Grade 3: somnolent, stuporous, place-disoriented, hyperactive reflexes, rigidity, slower waves.
  Grade 4: unrousable coma, no personality/behavior, decerebrate, slow 2-3 cps delta activity.
Time Frame: Day 1, Weeks 6, 12, 18, 24, 30, 36, and 48; and Extension Months 3, 6, 9, 12, and 15
Population: as for outcome 132
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Obeticholic Acid (OCA)
Number analyzed (Participants) | 12 | 10
Participants
  Baseline: Grade 0 | 7 | 7
  Baseline: Grade 1 or 2 | 5 | 3
  Baseline: Grade 3 or 4 | 0 | 0
  Day 1: Grade 0 | 8 | 8
  Day 1: Grade 1 or 2 | 4 | 2
  Day 1: Grade 3 or 4 | 0 | 0
  Week 6: number analyzed (Participants) | 9 | 9
  Week 6: Grade 0 | 6 | 6
  Week 6: Grade 1 or 2 | 3 | 3
  Week 6: Grade 3 or 4 | 0 | 0
  Week 12: number analyzed (Participants) | 6 | 7
  Week 12: Grade 0 | 4 | 5
  Week 12: Grade 1 or 2 | 2 | 2
  Week 12: Grade 3 or 4 | 0 | 0
  Week 18: number analyzed (Participants) | 8 | 8
  Week 18: Grade 0 | 6 | 7
  Week 18: Grade 1 or 2 | 2 | 1
  Week 18: Grade 3 or 4 | 0 | 0
  Week 24: number analyzed (Participants) | 6 | 6
  Week 24: Grade 0 | 6 | 5
  Week 24: Grade 1 or 2 | 0 | 1
  Week 24: Grade 3 or 4 | 0 | 0
  Week 30: number analyzed (Participants) | 6 | 6
  Week 30: Grade 0 | 5 | 5
  Week 30: Grade 1 or 2 | 1 | 1
  Week 30: Grade 3 or 4 | 0 | 0
  Week 36: number analyzed (Participants) | 6 | 6
  Week 36: Grade 0 | 6 | 5
  Week 36: Grade 1 or 2 | 0 | 1
  Week 36: Grade 3 or 4 | 0 | 0
  Week 48: number analyzed (Participants) | 6 | 6
  Week 48: Grade 0 | 5 | 5
  Week 48: Grade 1 or 2 | 1 | 1
  Week 48: Grade 3 or 4 | 0 | 0
  Extension Month 3: number analyzed (Participants) | 6 | 5
  Extension Month 3: Grade 0 | 5 | 4
  Extension Month 3: Grade 1 or 2 | 1 | 1
  Extension Month 3: Grade 3 or 4 | 0 | 0
  Extension Month 6: number analyzed (Participants) | 3 | 2
  Extension Month 6: Grade 0 | 3 | 1
  Extension Month 6: Grade 1 or 2 | 0 | 1
  Extension Month 6: Grade 3 or 4 | 0 | 0
  Extension Month 9: number analyzed (Participants) | 0 | 2
  Extension Month 9: Grade 0 | 0 | 1
  Extension Month 9: Grade 1 or 2 | 0 | 1
  Extension Month 9: Grade 3 or 4 | 0 | 0
  Extension Month 12: number analyzed (Participants) | 1 | 1
  Extension Month 12: Grade 0 | 1 | 0
  Extension Month 12: Grade 1 or 2 | 0 | 1
  Extension Month 12: Grade 3 or 4 | 0 | 0
  Extension Month 15: number analyzed (Participants) | 1 | 1
  Extension Month 15: Grade 0 | 1 | 0
  Extension Month 15: Grade 1 or 2 | 0 | 1
  Extension Month 15: Grade 3 or 4 | 0 | 0

140. Secondary Outcome: Change From Baseline in Total Bilirubin at Weeks 3, 6, 12, 18, 24, 30, 36, 42, and 48; and Extension Months 3, 6, 9, 12, and 15
Time Frame: Baseline, Weeks 3, 6, 12, 18, 24, 30, 36, 42, and 48; and Extension Months 3, 6, 9, 12, and 15
Population: as for outcome 132
Measure: Median (Inter-Quartile Range); unit: μmol/L
Arm/Group | Placebo | Obeticholic Acid (OCA)
Number analyzed (Participants) | 12 | 10
μmol/L
  Baseline | 45.38 [34.57 to 55.79] | 41.50 [19.00 to 106.88]
  Change at Week 3: number analyzed (Participants) | 11 | 10
  Change at Week 3 | 0.86 [-13.0 to 6.50] | -3.25 [-4.00 to 24.00]
  Change at Week 6: number analyzed (Participants) | 9 | 8
  Change at Week 6 | 3.00 [-1.50 to 5.99] | -2.14 [-3.43 to 26.75]
  Change at Week 12: number analyzed (Participants) | 7 | 7
  Change at Week 12 | 0.86 [-4.28 to 9.00] | -1.71 [-6.00 to 17.96]
  Change at Week 18: number analyzed (Participants) | 8 | 8
  Change at Week 18 | 1.08 [-4.70 to 16.05] | -4.03 [-9.00 to 3.21]
  Change at Week 24: number analyzed (Participants) | 5 | 7
  Change at Week 24 | 2.67 [-1.50 to 20.40] | -3.50 [-10.00 to 1.71]
  Change at Week 30: number analyzed (Participants) | 6 | 6
  Change at Week 30 | 2.08 [-2.57 to 31.34] | -8.49 [-9.00 to -5.50]
  Change at Week 36: number analyzed (Participants) | 6 | 6
  Change at Week 36 | 4.25 [-11.12 to 9.67] | -3.53 [-7.00 to 3.42]
  Change at Week 42: number analyzed (Participants) | 6 | 7
  Change at Week 42 | 6.58 [-7.70 to 12.00] | 1.71 [-2.85 to 6.00]
  Change at Week 48: number analyzed (Participants) | 6 | 6
  Change at Week 48 | 6.25 [-2.57 to 23.67] | -3.75 [-6.27 to -0.57]
  Change at Extension Month 3: number analyzed (Participants) | 6 | 5
  Change at Extension Month 3 | 2.25 [0.86 to 60.67] | 0.50 [-16.00 to 0.57]
  Change at Extension Month 6: number analyzed (Participants) | 3 | 2
  Change at Extension Month 6 | -1.50 [-12.83 to 21.38] | -0.22 [-1.00 to 0.57]
  Change at Extension Month 9: number analyzed (Participants) | 0 | 2
  Change at Extension Month 9 |  | -7.86 [-18.00 to 2.28]
  Change at Extension Month 12: number analyzed (Participants) | 1 | 1
  Change at Extension Month 12 | -14.54 [-14.54 to -14.54] | 9.12 [9.12 to 9.12]
  Change at Extension Month 15: number analyzed (Participants) | 1 | 1
  Change at Extension Month 15 | -12.83 [-12.83 to -12.83] | 24.51 [24.51 to 24.51]

141. Secondary Outcome: Change From Baseline in Direct Bilirubin at Weeks 3, 6, 12, 18, 24, 30, 36, 42, and 48; and Extension Months 3, 6, 9, 12, and 15
Time Frame: Baseline, Weeks 3, 6, 12, 18, 24, 30, 36, 42, and 48; and Extension Months 3, 6, 9, 12, and 15
Population: as for outcome 132
Measure: Median (Inter-Quartile Range); unit: μmol/L
Arm/Group | Placebo | Obeticholic Acid (OCA)
Number analyzed (Participants) | 12 | 10
μmol/L
  Baseline | 21.58 [15.37 to 37.18] | 25.50 [8.00 to 76.00]
  Change at Week 3: number analyzed (Participants) | 11 | 10
  Change at Week 3 | 0.00 [-6.04 to 1.50] | -1.07 [-1.50 to 15.00]
  Change at Week 6: number analyzed (Participants) | 8 | 8
  Change at Week 6 | 2.53 [0.00 to 7.25] | -1.32 [-4.61 to 18.50]
  Change at Week 12: number analyzed (Participants) | 7 | 7
  Change at Week 12 | 4.28 [0.00 to 12.50] | -1.14 [-3.00 to 1.71]
  Change at Week 18: number analyzed (Participants) | 8 | 8
  Change at Week 18 | 2.99 [0.50 to 14.20] | -1.82 [-3.25 to 2.00]
  Change at Week 24: number analyzed (Participants) | 5 | 6
  Change at Week 24 | 1.00 [-1.00 to 15.00] | -1.75 [-2.85 to 0.00]
  Change at Week 30: number analyzed (Participants) | 6 | 5
  Change at Week 30 | 0.93 [-1.00 to 6.10] | -2.50 [-4.00 to -1.71]
  Change at Week 36: number analyzed (Participants) | 6 | 6
  Change at Week 36 | 0.00 [-4.28 to 3.37] | -1.57 [-2.50 to 0.00]
  Change at Week 42: number analyzed (Participants) | 6 | 7
  Change at Week 42 | 2.50 [-2.57 to 9.37] | -1.71 [-2.66 to 1.50]
  Change at Week 48: number analyzed (Participants) | 6 | 6
  Change at Week 48 | 3.61 [-1.00 to 15.00] | -2.36 [-6.08 to -1.14]
  Change at Extension Month 3: number analyzed (Participants) | 5 | 5
  Change at Extension Month 3 | 3.37 [0.00 to 4.28] | -2.00 [-15.00 to 1.50]
  Change at Extension Month 6: number analyzed (Participants) | 3 | 2
  Change at Extension Month 6 | 0.00 [-5.99 to 19.67] | -1.00 [-6.00 to 3.99]
  Change at Extension Month 9: number analyzed (Participants) | 0 | 2
  Change at Extension Month 9 |  | -3.79 [-15.00 to 7.41]
  Change at Extension Month 12: number analyzed (Participants) | 1 | 1
  Change at Extension Month 12 | -9.41 [-9.41 to -9.41] | 7.41 [7.41 to 7.41]
  Change at Extension Month 15: number analyzed (Participants) | 1 | 1
  Change at Extension Month 15 | -5.99 [-5.99 to -5.99] | 12.54 [12.54 to 12.54]

142. Secondary Outcome: Change From Baseline in Alkaline Phosphatase at Weeks 3, 6, 12, 18, 24, 30, 36, 42, and 48; and Extension Months 3, 6, 9, 12, and 15
Time Frame: Baseline, Weeks 3, 6, 12, 18, 24, 30, 36, 42, and 48; and Extension Months 3, 6, 9, 12, and 15
Population: as for outcome 132
Measure: Median (Inter-Quartile Range); unit: unit per liter (U/L)
Arm/Group | Placebo | Obeticholic Acid (OCA)
Number analyzed (Participants) | 12 | 10
unit per liter (U/L)
  Baseline | 216.0 [144.5 to 290.0] | 267.5 [151.0 to 381.0]
  Change at Week 3: number analyzed (Participants) | 11 | 10
  Change at Week 3 | -21.0 [-48.0 to 6.0] | -9.0 [-48.0 to 0.0]
  Change at Week 6: number analyzed (Participants) | 9 | 9
  Change at Week 6 | -7.0 [-22.0 to 19.0] | 5.0 [-12.0 to 15.0]
  Change at Week 12: number analyzed (Participants) | 7 | 7
  Change at Week 12 | -1.0 [-54.0 to 12.0] | -17.0 [-32.0 to 6.0]
  Change at Week 18: number analyzed (Participants) | 8 | 8
  Change at Week 18 | -20.5 [-35.5 to 16.5] | -4.5 [-37.5 to 1.5]
  Change at Week 24: number analyzed (Participants) | 5 | 7
  Change at Week 24 | -30.0 [-66.0 to 16.0] | -5.0 [-100.0 to 4.0]
  Change at Week 30: number analyzed (Participants) | 6 | 6
  Change at Week 30 | -34.5 [-76.0 to -19.0] | -20.0 [-33.0 to -7.0]
  Change at Week 36: number analyzed (Participants) | 6 | 8
  Change at Week 36 | -26.0 [-64.0 to -6.0] | -4.0 [-89.5 to 4.0]
  Change at Week 42: number analyzed (Participants) | 6 | 7
  Change at Week 42 | -24.0 [-45.0 to -17.0] | 5.0 [-87.0 to 9.0]
  Change at Week 48: number analyzed (Participants) | 6 | 5
  Change at Week 48 | -29.0 [-63.0 to -17.0] | 8.0 [-3.0 to 13.0]
  Change at Extension Month 3: number analyzed (Participants) | 6 | 5
  Change at Extension Month 3 | -24.0 [-48.0 to -7.0] | 10.0 [-14.0 to 26.0]
  Change at Extension Month 6: number analyzed (Participants) | 3 | 2
  Change at Extension Month 6 | 6.0 [-33.0 to 7.0] | -46.0 [-133.0 to 41.0]
  Change at Extension Month 9: number analyzed (Participants) | 0 | 2
  Change at Extension Month 9 |  | -66.5 [-148.0 to 15.0]
  Change at Extension Month 12: number analyzed (Participants) | 1 | 1
  Change at Extension Month 12 | -72.0 [-72.0 to -72.0] | 122.0 [122.0 to 122.0]
  Change at Extension Month 15: number analyzed (Participants) | 1 | 1
  Change at Extension Month 15 | -83.0 [-83.0 to -83.0] | 10.0 [10.0 to 10.0]

143. Secondary Outcome: Change From Baseline in Alanine Aminotransferase at Weeks 3, 6, 12, 18, 24, 30, 36, 42, and 48; and Extension Months 3, 6, 9, 12, and 15
Time Frame: Baseline, Weeks 3, 6, 12, 18, 24, 30, 36, 42, and 48; and Extension Months 3, 6, 9, 12, and 15
Population: as for outcome 132
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | Placebo | Obeticholic Acid (OCA)
Number analyzed (Participants) | 12 | 10
U/L
  Baseline | 47.5 [31.0 to 60.5] | 38.0 [27.0 to 56.0]
  Change at Week 3: number analyzed (Participants) | 11 | 10
  Change at Week 3 | -5.0 [-9.0 to -1.0] | -2.0 [-9.0 to 1.0]
  Change at Week 6: number analyzed (Participants) | 9 | 8
  Change at Week 6 | -5.0 [-9.0 to 1.0] | 2.5 [-1.0 to 12.5]
  Change at Week 12: number analyzed (Participants) | 7 | 7
  Change at Week 12 | 1.0 [-9.0 to 5.0] | 10.0 [1.0 to 19.0]
  Change at Week 18: number analyzed (Participants) | 8 | 8
  Change at Week 18 | -6.5 [-12.5 to -3.5] | -0.5 [-5.0 to 1.5]
  Change at Week 24: number analyzed (Participants) | 5 | 6
  Change at Week 24 | -4.0 [-5.0 to 4.0] | -4.0 [-8.0 to 3.0]
  Change at Week 30: number analyzed (Participants) | 6 | 6
  Change at Week 30 | -6.0 [-12.0 to 3.0] | 1.5 [-2.0 to 3.0]
  Change at Week 36: number analyzed (Participants) | 6 | 7
  Change at Week 36 | 11.5 [-6.0 to 24.0] | -3.0 [-5.0 to 5.0]
  Change at Week 42: number analyzed (Participants) | 6 | 7
  Change at Week 42 | -9.0 [-12.0 to -3.0] | -1.0 [-6.0 to 1.0]
  Change at Week 48: number analyzed (Participants) | 6 | 6
  Change at Week 48 | -6.0 [-7.0 to -2.0] | 1.0 [-1.0 to 2.0]
  Change at Extension Month 3: number analyzed (Participants) | 6 | 5
  Change at Extension Month 3 | -8.0 [-12.0 to -3.0] | -1.0 [-7.0 to 7.0]
  Change at Extension Month 6: number analyzed (Participants) | 3 | 2
  Change at Extension Month 6 | -12.0 [-27.0 to -1.0] | -1.5 [-6.0 to 3.0]
  Change at Extension Month 9: number analyzed (Participants) | 0 | 2
  Change at Extension Month 9 |  | -6.0 [-11.0 to -1.0]
  Change at Extension Month 12: number analyzed (Participants) | 1 | 1
  Change at Extension Month 12 | -34.0 [-34.0 to -34.0] | -2.0 [-2.0 to -2.0]
  Change at Extension Month 15: number analyzed (Participants) | 1 | 1
  Change at Extension Month 15 | -32.0 [-32.0 to -32.0] | 1.0 [1.0 to 1.0]

144. Secondary Outcome: Change From Baseline in Aspartate Aminotransferase at Weeks 3, 6, 12, 18, 24, 30, 36, 42, and 48; and Extension Months 3, 6, 9, 12, and 15
Time Frame: Baseline, Weeks 3, 6, 12, 18, 24, 30, 36, 42, and 48; and Extension Months 3, 6, 9, 12, and 15
Population: as for outcome 132
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | Placebo | Obeticholic Acid (OCA)
Number analyzed (Participants) | 12 | 10
U/L
  Baseline | 60.0 [45.5 to 95.5] | 65.5 [46.0 to 104.0]
  Change at Week 3: number analyzed (Participants) | 11 | 10
  Change at Week 3 | -4.0 [-11.0 to 3.0] | -1.0 [-13.0 to 6.0]
  Change at Week 6: number analyzed (Participants) | 8 | 8
  Change at Week 6 | -4.0 [-12.0 to 0.5] | 10.5 [-3.5 to 23.5]
  Change at Week 12: number analyzed (Participants) | 7 | 7
  Change at Week 12 | 0.0 [-5.0 to 19.0] | 18.0 [-3.0 to 29.0]
  Change at Week 18: number analyzed (Participants) | 8 | 8
  Change at Week 18 | -1.5 [-7.5 to 5.5] | -5.0 [-10.5 to 4.5]
  Change at Week 24: number analyzed (Participants) | 5 | 6
  Change at Week 24 | -7.0 [-13.0 to -2.0] | -2.0 [-7.0 to 1.0]
  Change at Week 30: number analyzed (Participants) | 6 | 6
  Change at Week 30 | -10.0 [-12.0 to -3.0] | 1.0 [-2.0 to 9.0]
  Change at Week 36: number analyzed (Participants) | 6 | 7
  Change at Week 36 | 19.5 [-10.0 to 34.0] | 2.0 [-4.0 to 15.0]
  Change at Week 42: number analyzed (Participants) | 6 | 7
  Change at Week 42 | -3.5 [-14.0 to 8.0] | 1.0 [-2.0 to 39.0]
  Change at Week 48: number analyzed (Participants) | 6 | 6
  Change at Week 48 | -12.0 [-22.0 to 7.0] | 0.5 [-15.0 to 20.0]
  Change at Extension Month 3: number analyzed (Participants) | 6 | 5
  Change at Extension Month 3 | -6.5 [-11.0 to 6.0] | -12.0 [-15.0 to 6.0]
  Change at Extension Month 6: number analyzed (Participants) | 3 | 2
  Change at Extension Month 6 | -16.0 [-32.0 to 1.0] | -0.5 [-21.0 to 20.0]
  Change at Extension Month 9: number analyzed (Participants) | 0 | 2
  Change at Extension Month 9 |  | -8.5 [-33.0 to 16.0]
  Change at Extension Month 12: number analyzed (Participants) | 1 | 1
  Change at Extension Month 12 | -33.0 [-33.0 to -33.0] | 19.0 [19.0 to 19.0]
  Change at Extension Month 15: number analyzed (Participants) | 1 | 1
  Change at Extension Month 15 | -34.0 [-34.0 to -34.0] | 16.0 [16.0 to 16.0]

145. Secondary Outcome: Change From Baseline in Gamma Glutamyl Transferase at Weeks 3, 6, 12, 18, 24, 30, 36, 42, and 48; and Extension Months 3, 6, 9, 12, and 15
Time Frame: Baseline, Weeks 3, 6, 12, 18, 24, 30, 36, 42, and 48; and Extension Months 3, 6, 9, 12, and 15
Population: as for outcome 132
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | Placebo | Obeticholic Acid (OCA)
Number analyzed (Participants) | 12 | 10
U/L
  Baseline | 98.0 [36.0 to 152.0] | 103.0 [53.0 to 191.0]
  Change at Week 3: number analyzed (Participants) | 10 | 10
  Change at Week 3 | -12.5 [-27.0 to -2.0] | -13.5 [-54.0 to -1.0]
  Change at Week 6: number analyzed (Participants) | 9 | 9
  Change at Week 6 | -11.0 [-28.0 to -3.0] | 0.0 [-31.0 to 4.0]
  Change at Week 12: number analyzed (Participants) | 7 | 7
  Change at Week 12 | -13.0 [-32.0 to -3.0] | -2.0 [-44.0 to 7.0]
  Change at Week 18: number analyzed (Participants) | 8 | 8
  Change at Week 18 | -9.5 [-28.0 to -0.5] | -3.5 [-38.5 to 1.5]
  Change at Week 24: number analyzed (Participants) | 5 | 7
  Change at Week 24 | 8.0 [-37.0 to 25.0] | -14.0 [-70.0 to -5.0]
  Change at Week 30: number analyzed (Participants) | 5 | 6
  Change at Week 30 | -9.0 [-22.0 to -5.0] | -12.5 [-27.0 to 5.0]
  Change at Week 36: number analyzed (Participants) | 6 | 8
  Change at Week 36 | -5.5 [-12.0 to 24.0] | -10.5 [-90.0 to 4.5]
  Change at Week 42: number analyzed (Participants) | 6 | 7
  Change at Week 42 | -12.0 [-26.0 to 5.0] | -4.0 [-154.0 to 17.0]
  Change at Week 48: number analyzed (Participants) | 6 | 6
  Change at Week 48 | -9.0 [-21.0 to -6.0] | -15.0 [-112.0 to 9.0]
  Change at Extension Month 3: number analyzed (Participants) | 6 | 5
  Change at Extension Month 3 | -9.5 [-48.0 to 1.0] | 9.0 [-14.0 to 22.0]
  Change at Extension Month 6: number analyzed (Participants) | 3 | 2
  Change at Extension Month 6 | -10.0 [-35.0 to -9.0] | -58.5 [-137.0 to 20.0]
  Change at Extension Month 9: number analyzed (Participants) | 0 | 2
  Change at Extension Month 9 |  | -57.0 [-128.0 to 14.0]
  Change at Extension Month 12: number analyzed (Participants) | 1 | 1
  Change at Extension Month 12 | -74.0 [-74.0 to -74.0] | 8.0 [8.0 to 8.0]
  Change at Extension Month 15: number analyzed (Participants) | 1 | 1
  Change at Extension Month 15 | -63.0 [-63.0 to -63.0] | 2.0 [2.0 to 2.0]

146. Secondary Outcome: Change From Baseline in Prothrombin INR at Weeks 3, 6, 12, 18, 24, 30, 36, 42, and 48; and Extension Months 3, 6, 9, 12, and 15
Time Frame: Baseline, Weeks 3, 6, 12, 18, 24, 30, 36, 42, and 48; and Extension Months 3, 6, 9, 12, and 15
Population: as for outcome 132
Measure: Median (Inter-Quartile Range); unit: INR
Arm/Group | Placebo | Obeticholic Acid (OCA)
Number analyzed (Participants) | 12 | 10
INR
  Baseline | 1.15 [1.10 to 1.20] | 1.23 [1.10 to 1.30]
  Change at Week 3: number analyzed (Participants) | 11 | 10
  Change at Week 3 | 0.00 [0.00 to 0.10] | 0.00 [0.00 to 0.10]
  Change at Week 6: number analyzed (Participants) | 9 | 9
  Change at Week 6 | 0.00 [-0.03 to 0.00] | 0.00 [-0.05 to 0.00]
  Change at Week 12: number analyzed (Participants) | 6 | 7
  Change at Week 12 | 0.08 [0.00 to 0.15] | -0.05 [-0.10 to 0.00]
  Change at Week 18: number analyzed (Participants) | 8 | 8
  Change at Week 18 | 0.09 [0.00 to 0.10] | -0.05 [-0.13 to 0.05]
  Change at Week 24: number analyzed (Participants) | 4 | 5
  Change at Week 24 | 0.03 [-0.02 to 0.08] | -0.05 [-0.10 to 0.05]
  Change at Week 30: number analyzed (Participants) | 6 | 6
  Change at Week 30 | 0.03 [-0.03 to 0.10] | 0.00 [-0.10 to 0.00]
  Change at Week 36: number analyzed (Participants) | 6 | 8
  Change at Week 36 | 0.05 [0.00 to 0.10] | -0.10 [-0.18 to 0.03]
  Change at Week 42: number analyzed (Participants) | 6 | 7
  Change at Week 42 | 0.05 [0.00 to 0.07] | 0.00 [-0.10 to 0.05]
  Change at Week 48: number analyzed (Participants) | 6 | 5
  Change at Week 48 | 0.00 [-0.03 to 0.05] | -0.10 [-0.15 to 0.00]
  Change at Extension Month 3: number analyzed (Participants) | 6 | 5
  Change at Extension Month 3 | 0.06 [0.00 to 0.10] | -0.10 [-0.10 to -0.10]
  Change at Extension Month 6: number analyzed (Participants) | 3 | 2
  Change at Extension Month 6 | 0.05 [-0.10 to 0.15] | -0.05 [-0.10 to 0.00]
  Change at Extension Month 9: number analyzed (Participants) | 1 | 2
  Change at Extension Month 9 | 0.15 [0.15 to 0.15] | 0.00 [0.00 to 0.00]
  Change at Extension Month 12: number analyzed (Participants) | 1 | 1
  Change at Extension Month 12 | 0.05 [0.05 to 0.05] | 0.10 [0.10 to 0.10]
  Change at Extension Month 15: number analyzed (Participants) | 1 | 0
  Change at Extension Month 15 | 0.05 [0.05 to 0.05] |

147. Secondary Outcome: Change From Baseline in Creatinine at Weeks 3, 6, 12, 18, 24, 30, 36, 42, and 48; and Extension Months 3, 6, 9, 12, and 15
Time Frame: Baseline, Weeks 3, 6, 12, 18, 24, 30, 36, 42, and 48; and Extension Months 3, 6, 9, 12, and 15
Population: as for outcome 132
Measure: Median (Inter-Quartile Range); unit: µmol/L
Arm/Group | Placebo | Obeticholic Acid (OCA)
Number analyzed (Participants) | 12 | 10
µmol/L
  Baseline | 60.000 [51.000 to 96.732] | 60.172 [55.000 to 95.472]
  Change at Week 3: number analyzed (Participants) | 11 | 10
  Change at Week 3 | 0.884 [-3.000 to 5.000] | -0.308 [-2.000 to 1.768]
  Change at Week 6: number analyzed (Participants) | 9 | 9
  Change at Week 6 | 5.000 [0.388 to 5.746] | 0.884 [-1.000 to 4.000]
  Change at Week 12: number analyzed (Participants) | 7 | 7
  Change at Week 12 | -0.496 [-4.000 to 13.500] | 2.500 [-1.000 to 5.000]
  Change at Week 18: number analyzed (Participants) | 8 | 8
  Change at Week 18 | -2.431 [-4.958 to 7.250] | 0.942 [-6.170 to 5.036]
  Change at Week 24: number analyzed (Participants) | 5 | 7
  Change at Week 24 | -1.000 [-4.000 to -0.496] | -2.652 [-11.492 to 5.000]
  Change at Week 30: number analyzed (Participants) | 6 | 6
  Change at Week 30 | -0.663 [-4.032 to 1.768] | -2.250 [-6.188 to 3.000]
  Change at Week 36: number analyzed (Participants) | 6 | 8
  Change at Week 36 | 1.500 [-1.326 to 7.000] | 2.466 [-1.960 to 33.586]
  Change at Week 42: number analyzed (Participants) | 6 | 7
  Change at Week 42 | 2.000 [-1.326 to 4.000] | 6.236 [-2.652 to 28.000]
  Change at Week 48: number analyzed (Participants) | 6 | 6
  Change at Week 48 | 2.221 [-3.536 to 6.000] | 0.466 [-3.000 to 20.000]
  Change at Extension Month 3: number analyzed (Participants) | 6 | 5
  Change at Extension Month 3 | 3.884 [0.000 to 6.630] | 0.000 [-1.500 to 12.000]
  Change at Extension Month 6: number analyzed (Participants) | 3 | 2
  Change at Extension Month 6 | 2.652 [-4.000 to 12.818] | 4.648 [-7.500 to 16.796]
  Change at Extension Month 9: number analyzed (Participants) | 0 | 2
  Change at Extension Month 9 |  | 15.068 [4.500 to 25.636]
  Change at Extension Month 12: number analyzed (Participants) | 1 | 1
  Change at Extension Month 12 | 10.608 [10.608 to 10.608] | 27.404 [27.404 to 27.404]
  Change at Extension Month 15: number analyzed (Participants) | 1 | 1
  Change at Extension Month 15 | 4.420 [4.420 to 4.420] | 29.172 [29.172 to 29.172]

148. Secondary Outcome: Change From Baseline in Albumin at Weeks 3, 6, 12, 18, 24, 30, 36, 42, and 48; and Extension Months 3, 6, 9, 12, and 15
Time Frame: Baseline, Weeks 3, 6, 12, 18, 24, 30, 36, 42, and 48; and Extension Months 3, 6, 9, 12, and 15
Population: as for outcome 132
Measure: Median (Inter-Quartile Range); unit: g/L
Arm/Group | Placebo | Obeticholic Acid (OCA)
Number analyzed (Participants) | 12 | 10
g/L
  Baseline | 34.50 [33.00 to 36.75] | 33.00 [30.00 to 36.50]
  Change at Week 3: number analyzed (Participants) | 10 | 10
  Change at Week 3 | -2.25 [-2.50 to -1.00] | -0.50 [-1.70 to 0.00]
  Change at Week 6: number analyzed (Participants) | 9 | 9
  Change at Week 6 | -1.00 [-3.00 to 0.00] | 0.00 [-1.00 to 1.30]
  Change at Week 12: number analyzed (Participants) | 7 | 7
  Change at Week 12 | -2.00 [-4.00 to -1.50] | -0.70 [-1.00 to 1.50]
  Change at Week 18: number analyzed (Participants) | 8 | 8
  Change at Week 18 | -4.25 [-5.00 to -1.50] | 0.00 [-1.60 to 0.50]
  Change at Week 24: number analyzed (Participants) | 5 | 7
  Change at Week 24 | -2.50 [-4.00 to -1.00] | -2.50 [-2.70 to 1.00]
  Change at Week 30: number analyzed (Participants) | 6 | 6
  Change at Week 30 | -2.50 [-4.00 to -2.00] | 0.15 [-1.50 to 1.00]
  Change at Week 36: number analyzed (Participants) | 6 | 8
  Change at Week 36 | -2.00 [-3.00 to -2.00] | 0.50 [-2.35 to 2.25]
  Change at Week 42: number analyzed (Participants) | 6 | 7
  Change at Week 42 | -1.25 [-4.00 to 0.00] | -0.70 [-1.00 to 2.00]
  Change at Week 48: number analyzed (Participants) | 6 | 6
  Change at Week 48 | -0.50 [-2.00 to 1.00] | 0.50 [-4.70 to 1.00]
  Change at Extension Month 3: number analyzed (Participants) | 6 | 5
  Change at Extension Month 3 | -2.50 [-3.00 to -1.00] | 1.00 [-2.70 to 2.50]
  Change at Extension Month 6: number analyzed (Participants) | 3 | 2
  Change at Extension Month 6 | -2.00 [-3.00 to -1.00] | -0.35 [-1.70 to 1.00]
  Change at Extension Month 9: number analyzed (Participants) | 0 | 2
  Change at Extension Month 9 |  | -1.35 [-3.70 to 1.00]
  Change at Extension Month 12: number analyzed (Participants) | 1 | 1
  Change at Extension Month 12 | -1.00 [-1.00 to -1.00] | -2.70 [-2.70 to -2.70]
  Change at Extension Month 15: number analyzed (Participants) | 1 | 1
  Change at Extension Month 15 | -1.00 [-1.00 to -1.00] | -11.70 [-11.70 to -11.70]

149. Secondary Outcome: Change From Baseline in Platelets at Weeks 3, 6, 12, 18, 24, 30, 36, 42, and 48; and Extension Months 3, 6, 9, 12, and 15
Time Frame: Baseline, Weeks 3, 6, 12, 18, 24, 30, 36, 42, and 48; and Extension Months 3, 6, 9, 12, and 15
Population: as for outcome 132
Measure: Median (Inter-Quartile Range); unit: 10^9/L
Arm/Group | Placebo | Obeticholic Acid (OCA)
Number analyzed (Participants) | 11 | 9
10^9/L
  Baseline | 141.5 [80.0 to 160.5] | 132.5 [84.5 to 158.5]
  Change at Week 3: number analyzed (Participants) | 10 | 9
  Change at Week 3 | -6.2 [-21.0 to -3.0] | -7.5 [-12.0 to 8.5]
  Change at Week 6: number analyzed (Participants) | 8 | 6
  Change at Week 6 | -12.0 [-28.8 to -2.3] | 15.0 [1.0 to 26.5]
  Change at Week 12: number analyzed (Participants) | 6 | 5
  Change at Week 12 | -10.5 [-31.0 to 7.5] | -15.0 [-15.0 to -1.5]
  Change at Week 18: number analyzed (Participants) | 6 | 7
  Change at Week 18 | -15.0 [-21.9 to -8.5] | 7.5 [-10.0 to 38.5]
  Change at Week 24: number analyzed (Participants) | 5 | 6
  Change at Week 24 | 4.5 [-14.4 to 17.0] | -1.5 [-25.0 to 25.5]
  Change at Week 30: number analyzed (Participants) | 6 | 5
  Change at Week 30 | -11.4 [-23.5 to 15.0] | -5.5 [-9.0 to 6.5]
  Change at Week 36: number analyzed (Participants) | 6 | 6
  Change at Week 36 | -16.5 [-20.5 to -12.0] | 9.8 [-6.5 to 39.5]
  Change at Week 42: number analyzed (Participants) | 6 | 6
  Change at Week 42 | -16.2 [-37.5 to -10.0] | 9.0 [6.5 to 11.0]
  Change at Week 48: number analyzed (Participants) | 5 | 5
  Change at Week 48 | 4.0 [-41.5 to 23.0] | -9.0 [-11.5 to 14.5]
  Change at Extension Month 3: number analyzed (Participants) | 6 | 5
  Change at Extension Month 3 | -5.0 [-24.0 to 16.5] | -11.5 [-24.0 to -8.5]
  Change at Extension Month 6: number analyzed (Participants) | 3 | 1
  Change at Extension Month 6 | 48.5 [14.0 to 78.0] | -0.5 [-0.5 to -0.5]
  Change at Extension Month 9: number analyzed (Participants) | 0 | 2
  Change at Extension Month 9 |  | -4.5 [-5.5 to -3.5]
  Change at Extension Month 12: number analyzed (Participants) | 1 | 1
  Change at Extension Month 12 | -2.0 [-2.0 to -2.0] | -3.5 [-3.5 to -3.5]
  Change at Extension Month 15: number analyzed (Participants) | 1 | 1
  Change at Extension Month 15 | -9.0 [-9.0 to -9.0] | -22.5 [-22.5 to -22.5]

150. Secondary Outcome: Change From Baseline in Total Bile Acids Concentration at Weeks 6, 12, 18, 24, 30, 36, and 48; and Extension Month 3
Description: Total bile acids (micromole [μM]) = total ursodeoxycholic acid (unconjugated, glyco-conjugate, tauro-conjugate) in μM + total chenodeoxycholic acid (unconjugated, glyco-conjugate, tauro-conjugate) in μM + total deoxycholic acid (unconjugated, glyco-conjugate, tauro-conjugate) in μM + total cholic acid (unconjugated, glyco-conjugate, tauro-conjugate) in μM + total lithocholic acid (unconjugated, glyco-conjugate, tauro-conjugate) in μM.
Time Frame: Baseline, Weeks 6, 12, 18, 24, 30, 36, and 48; and Extension Month 3
Population: as for outcome 132
Measure: Median (Inter-Quartile Range); unit: μM
Arm/Group | Placebo | Obeticholic Acid (OCA)
Number analyzed (Participants) | 11 | 10
μM
  Baseline | 149 [90.3 to 307] | 127 [65.3 to 176]
  Change at Week 6: number analyzed (Participants) | 7 | 8
  Change at Week 6 | 16.3 [-7.68 to 37.4] | 8.09 [-15.9 to 37.1]
  Change at Week 12: number analyzed (Participants) | 6 | 6
  Change at Week 12 | 0.863 [-21.0 to 88.4] | 5.55 [-58.4 to 13.7]
  Change at Week 18: number analyzed (Participants) | 11 | 7
  Change at Week 18 | 17.7 [-56.0 to 160] | 12.8 [-169 to 36.0]
  Change at Week 24: number analyzed (Participants) | 4 | 4
  Change at Week 24 | 3.29 [-76.6 to 30.6] | -3.14 [-14.5 to 21.3]
  Change at Week 30: number analyzed (Participants) | 4 | 6
  Change at Week 30 | 26.0 [-56.0 to 98.5] | 16.1 [-7.06 to 38.7]
  Change at Week 36: number analyzed (Participants) | 5 | 10
  Change at Week 36 | -15.2 [-79.4 to 10.0] | -1.54 [-22.9 to 24.6]
  Change at Week 48: number analyzed (Participants) | 4 | 5
  Change at Week 48 | 63.2 [16.7 to 132] | 0.876 [-4.07 to 19.5]
  Change at Extension Month 3: number analyzed (Participants) | 0 | 1
  Change at Extension Month 3 |  | -32.9 [-32.9 to -32.9]

151. Secondary Outcome: Change From Baseline in Total Endogenous Bile Acids Concentration at Weeks 6, 12, 18, 24, 30, 36, and 48; and Extension Month 3
Description: Total endogenous bile acids (μM) = total chenodeoxycholic acid (unconjugated, glyco-conjugate, tauro-conjugate) in μM + total deoxycholic acid (unconjugated, glyco-conjugate, tauro-conjugate) in μM + total cholic acid (unconjugated, glyco-conjugate, tauro-conjugate) in μM + total lithocholic acid (unconjugated, glyco-conjugate, tauro-conjugate) in μM.
Time Frame: Baseline, Weeks 6, 12, 18, 24, 30, 36, and 48; and Extension Month 3
Population: as for outcome 132
Measure: Median (Inter-Quartile Range); unit: μM
Arm/Group | Placebo | Obeticholic Acid (OCA)
Number analyzed (Participants) | 11 | 10
μM
  Baseline | 64.7 [29.4 to 75.2] | 42.1 [18.6 to 69.6]
  Change at Week 6: number analyzed (Participants) | 7 | 9
  Change at Week 6 | -4.98 [-6.88 to 36.2] | 3.58 [-5.64 to 14.0]
  Change at Week 12: number analyzed (Participants) | 6 | 6
  Change at Week 12 | -3.97 [-13.3 to 63.9] | 1.46 [-5.43 to 4.81]
  Change at Week 18: number analyzed (Participants) | 11 | 7
  Change at Week 18 | -5.00 [-20.2 to 51.0] | 3.98 [-18.3 to 7.21]
  Change at Week 24: number analyzed (Participants) | 4 | 6
  Change at Week 24 | -6.76 [-18.5 to -1.25] | 3.18 [-2.53 to 15.2]
  Change at Week 30: number analyzed (Participants) | 5 | 6
  Change at Week 30 | 6.74 [-6.22 to 7.44] | 1.47 [-3.87 to 13.6]
  Change at Week 36: number analyzed (Participants) | 6 | 8
  Change at Week 36 | -5.74 [-24.9 to -0.576] | -2.69 [-14.4 to 9.66]
  Change at Week 48: number analyzed (Participants) | 6 | 6
  Change at Week 48 | 10.9 [6.32 to 19.8] | 4.18 [-2.08 to 9.82]
  Change at Extension Month 3: number analyzed (Participants) | 0 | 1
  Change at Extension Month 3 |  | -9.57 [-9.57 to -9.57]

152. Secondary Outcome: Change From Baseline in 7α-hydroxy-4-cholesten-3-one (C4) at Weeks 6, 12, 18, 24, 30, 36, and 48; and Extension Month 3
Time Frame: Baseline, Weeks 6, 12, 18, 24, 30, 36, and 48; and Extension Month 3
Population: as for outcome 132
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Placebo | Obeticholic Acid (OCA)
Number analyzed (Participants) | 11 | 10
ng/mL
  Baseline | 0.708 [0.372 to 5.16] | 0.814 [0.472 to 2.09]
  Change at Week 6: number analyzed (Participants) | 8 | 9
  Change at Week 6 | 0.0990 [-0.0445 to 0.296] | 0.0770 [-0.110 to 0.450]
  Change at Week 12: number analyzed (Participants) | 6 | 7
  Change at Week 12 | -0.0275 [-0.0690 to 0.156] | -0.289 [-1.31 to 0.0100]
  Change at Week 18: number analyzed (Participants) | 7 | 8
  Change at Week 18 | -0.0470 [-0.278 to 0.205] | -0.267 [-0.965 to 8.05]
  Change at Week 24: number analyzed (Participants) | 4 | 6
  Change at Week 24 | -0.00100 [-0.00700 to 0.692] | -0.141 [-1.67 to 1.07]
  Change at Week 30: number analyzed (Participants) | 5 | 6
  Change at Week 30 | 0.0890 [0.0500 to 0.355] | -0.386 [-1.77 to 2.50]
  Change at Week 36: number analyzed (Participants) | 6 | 8
  Change at Week 36 | 0.118 [-0.104 to 0.240] | -0.476 [-3.53 to 5.41]
  Change at Week 48: number analyzed (Participants) | 6 | 6
  Change at Week 48 | -0.170 [-0.491 to -0.0140] | -0.510 [-1.83 to 5.20]
  Change at Extension Month 3: number analyzed (Participants) | 0 | 1
  Change at Extension Month 3 |  | 1.36 [1.36 to 1.36]

153. Secondary Outcome: Change From Baseline in Fibroblast Growth Factor-19 (FGF-19) Concentrations at Weeks 6, 12, 18, 24, 30, 36, and 48; and Extension Month 3
Time Frame: Baseline, Weeks 6, 12, 18, 24, 30, 36, and 48; and Extension Month 3
Population: as for outcome 132
Measure: Median (Inter-Quartile Range); unit: picograms per milliliter (pg/mL)
Arm/Group | Placebo | Obeticholic Acid (OCA)
Number analyzed (Participants) | 11 | 10
picograms per milliliter (pg/mL)
  Baseline | 278 [105 to 618] | 163 [139 to 359]
  Change at Week 6: number analyzed (Participants) | 8 | 9
  Change at Week 6 | -50.7 [-142 to 33.0] | 26.0 [4.50 to 101]
  Change at Week 12: number analyzed (Participants) | 6 | 7
  Change at Week 12 | -14.0 [-220 to 19.0] | 119 [-25.6 to 174]
  Change at Week 18: number analyzed (Participants) | 7 | 8
  Change at Week 18 | -57.0 [-118 to 40.0] | 136 [-28.3 to 298]
  Change at Week 24: number analyzed (Participants) | 4 | 6
  Change at Week 24 | -33.0 [-152 to 402] | 16.6 [-24.0 to 219]
  Change at Week 30: number analyzed (Participants) | 5 | 6
  Change at Week 30 | -83.0 [-123 to 43.0] | 142 [-45.0 to 168]
  Change at Week 36: number analyzed (Participants) | 6 | 8
  Change at Week 36 | 26.0 [-34.0 to 102] | 15.0 [-97.4 to 201]
  Change at Week 48: number analyzed (Participants) | 6 | 6
  Change at Week 48 | -28.5 [-161 to 84.5] | 69.6 [8.00 to 145]
  Change at Extension Month 3: number analyzed (Participants) | 1 | 1
  Change at Extension Month 3 | -117 [-117 to -117] | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: Baseline up to approximately 3 years
Description: The Safety Population included all participants who received at least 1 dose of investigational product (OCA or placebo). Data were prespecified to be collected per randomization arm (OCA or placebo). Data at the separate dose levels are not available.
Arm/Group | Placebo | Obeticholic Acid (OCA)
All-Cause Mortality (participants affected / at risk) | 2/12 | 2/10
Serious Adverse Events (participants affected / at risk) | 9/12 | 7/10
Other Adverse Events (participants affected / at risk) | 10/12 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=12) | Obeticholic Acid (OCA) (N=10)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 3
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
COVID-19 (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Liver transplant (Surgical and medical procedures) | 1 | 0
Aortic aneurysm rupture (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=12) | Obeticholic Acid (OCA) (N=10)
Ascites (Gastrointestinal disorders) | 4 | 6
Abdominal distension (Gastrointestinal disorders) | 3 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 2 | 2
Vomiting (Gastrointestinal disorders) | 1 | 2
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0
Gastric antral vascular ectasia (Gastrointestinal disorders) | 1 | 0
Gastric polyps (Gastrointestinal disorders) | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0
Portal hypertensive gastropathy (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Varices oesophageal (Gastrointestinal disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 3
Pneumonia (Infections and infestations) | 0 | 2
Cytomegalovirus infection reactivation (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 0 | 1
Peritonitis bacterial (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 1 | 0
Fungal infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Fatigue (General disorders) | 1 | 2
Chest discomfort (General disorders) | 0 | 1
Disease progression (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 4 | 1
Asthenia (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 2
Balance disorder (Nervous system disorders) | 0 | 1
Burning sensation (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 1
Hepatic encephalopathy (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 1
Neuralgia (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 3
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 1
Palmar erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 3
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Limb mass (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 1
Blood urea increased (Investigations) | 0 | 1
Cardiac murmur (Investigations) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1
Thyroid mass (Endocrine disorders) | 0 | 1
Vitreous floaters (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 2 | 1
Joint injury (Injury, poisoning and procedural complications) | 2 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Breast pain (Reproductive system and breast disorders) | 1 | 0
Peripheral coldness (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 0
Haemorrhage (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators must wait 18 months after the study ends to publish their results and a multi-center publication must come first. The sponsor has a 45 day review period with the option to extend to an additional 90 days.

DOCUMENTS (2):
  • Study Protocol (2020-05-19): https://cdn.clinicaltrials.gov/large-docs/27/NCT03633227/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-27): https://cdn.clinicaltrials.gov/large-docs/27/NCT03633227/SAP_001.pdf